CLINICAL TRIAL: NCT03086460
Title: A Randomized, Double-blind, Placebo and Active-controlled, Incomplete Block Cross-over, Dose Ranging Study to Evaluate the Efficacy and Safety of 4 Doses of CHF 1531 pMDI (Formoterol Fumarate) in Asthmatic Subjects
Brief Title: A Dose Ranging Study With CHF 1531 in Subjects With Asthma (FLASH)
Acronym: FLASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CCD-05993AA3-03
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment A (Experimental): Treatment A, CHF 1531 pMDI:
  CHF 1531 pMDI 6 μg total daily dose (TDD):
  1 inhalation of CHF 1531 pMDI 3 μg/actuation plus 1 inhalation of CHF 1531 matched Placebo BID.
  Interventions: Drug: CHF 1531 pMDI
- Treatment B (Experimental): Treatment B, CHF 1531 pMDI:
  CHF 1531 pMDI 12 μg TDD:
  1 inhalation of CHF 1531 pMDI 6 μg/actuation plus 1 inhalation of CHF 1531 matched Placebo BID.
  Interventions: Drug: CHF 1531 pMDI
- Treatment C (Experimental): Treatment C, CHF 1531 pMDI:
  CHF 1531 pMDI 24 μg TDD: 2 inhalations of CHF 1531 pMDI 6 μg/actuation BID.
  Interventions: Drug: CHF 1531 pMDI
- Treatment D (Experimental): Treatment D, CHF 1531 pMDI
  CHF 1531 pMDI 48 μg TDD: 2 inhalations of CHF 1531 pMDI 12 μg/actuation BID.
  Interventions: Drug: CHF 1531 pMDI
- Treatment E (Experimental): Treatment E, Matched placebo
  Placebo: 2 inhalations of CHF 1531 pMDI matched Placebo BID.
  Interventions: Drug: Placebo pMDI
- Treatment F (Active Comparator): Treatment F, Formoterol fumarate inhalation solution (IS)
  Perforomist® IS (active comparator, open-label) 40 μg TDD: 1 inhalation, 20 μg/ 2 mL vial, 1 vial BID.
  Interventions: Drug: Formoterol Inhalation Solution

INTERVENTIONS:
Drug: CHF 1531 pMDI — Dose Response: Test one of five different doses of CHF 1531
  Arms: Treatment A; Treatment B; Treatment C; Treatment D
Drug: Formoterol Inhalation Solution — Active Control
  Other Names: PERFOROMIST® 20 μg/ 2 mL vial, 1 vial BID
  Arms: Treatment F
Drug: Placebo pMDI — Matched Placebo
  Arms: Treatment E

SUMMARY:
To evaluate the dose-response of different doses of CHF 1531 pressurized metered dose inhaler (pMDI) containing formoterol fumarate, on lung function and other clinical outcomes and to identify the optimal dose(s) with regard to benefit/ risk ratio for further development in the target subject population.

DETAILED DESCRIPTION:
This is a phase II, randomized, double-blind, placebo and active controlled dose-ranging, 6 arm incomplete block cross-over study to identify the optimal dose of CHF 1531 pMDI (containing formoterol fumarate), with regard to lung function and other clinical efficacy and safety outcome measures.

After a 2 week run-in period under rescue albuterol 'as needed' and background inhaled corticosteroid (ICS), subjects qualifying for the study were required to complete 4 treatment intervals of 2 weeks each, separated by 2 week wash-out intervals.

During each treatment interval, the subject were randomly assigned to take one of 5 double-blind study treatments twice daily (BID) i.e. one of 4 doses of CHF 1531 pMDI or a matching placebo or the open-label active control treatment (Perforomist® Inhalation Solution [IS]) also BID. During the entire study, all subjects concomitantly received ICS treatment with QVAR® inhaler (beclomethasone dipropionate 40 or 80 µg /actuation) twice daily at a dose that matches their pre-enrollment ICS and an albuterol inhaler to use as asthma rescue medication on 'as needed' basis. The subjects visited the study center every 2 weeks to undergo study procedures, and received a safety follow-up phone call one week after their last visit. In total, the study lasted 18 weeks and required 10 visits to the study center.

During the study, daily asthma symptoms, peak expiratory flow, rescue and background medication use, and compliance with the study medication were recorded in a subject diary. Treatment-Emergent Adverse Events (TEAEs) were assessed and recorded throughout the study. A full physical exam, routine hematology, blood chemistry, spirometry, vital signs measurement, 12-lead ECG, and pregnancy testing were performed before enrollment and at the end of the study. Furthermore, on Day 1 and 14 of each treatment interval, serial spirometry, 12-lead ECGs, blood pressure measurements (BP), serum potassium, and serum glucose were measured at the study center for up to 12 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 and ≤75 years who have signed an Informed Consent Form prior to initiation of any study-related procedure.
* A diagnosis of asthma as defined in the Global Initiative for Asthma (GINA) Report, 2016, documented for at least 1 year prior to screening.
* Poorly controlled or uncontrolled asthma evidenced by a score ≥1.5 on the Asthma Control Questionnaire 7 © (ACQ-7)
* A pre-bronchodilator Forced Expiratory Volume in the 1st Second ( FEV1) ≥60% and <85% of their predicted normal value, after appropriate washout from bronchodilators, at the screening and randomization visits
* Subjects with a positive response to a reversibility test at screening, defined as change in FEV1 (ΔFEV1) ≥12% and ≥200 mL over baseline within 30 minutes after inhaling 4 puffs of albuterol hydrofluoroalkane(HFA) 90 µg/actuation.
* Use of ICS (low/medium dose according to GINA Report, 2016) with or without a long-acting bronchodilator for 3 months (at a stable dose in the last 4 weeks) before screening visit.
* A cooperative attitude and ability to demonstrate correct use of the diary, peak flow meter, and pMDI inhaler.

Exclusion Criteria:

* Pregnant or lactating women and all women physiologically capable of becoming pregnant UNLESS they are willing to use a highly effective birth control methods
* Subjects who suffer from Chronic Obstructive Pulmonary Disease (COPD) as defined by the Global Strategy for Prevention, Diagnosis and Management of COPD (GOLD) Report, 2017, or are suspected of having Asthma COPD Overlap Syndrome (ACOS) as described in the GINA Report, 2016.
* Inability to carry out pulmonary function testing, to comply with study procedures or with study drug intake.
* Current smokers or ex-smokers (tobacco, vapor cigarettes, marijuana) with a smoking history of >10 pack-years or having stopped smoking one year or less prior to screening visit.
* History of life-threatening asthma, clinically significant uncontrolled disease or respiratory infection.
* An asthma exacerbation requiring oral/intravenous corticosteroids ≤ 30 days, intramuscular depot corticosteroid ≤3 months or hospitalization within 6 months prior to screening.
* Subjects with unresolved bacterial or viral respiratory tract, sinus, or middle ear infection affecting asthma status within 2 weeks prior to screening.
* Subjects who received a vaccination within 2 weeks prior to screening or during the run-in.
* Subjects with oral candidiasis at screening and at randomization.
* Subjects with any clinically significant, uncontrolled condition.
* Subjects with serum potassium levels <3.5 milliequivalents per litre (mEq/L) or (3.5 mmol/L) at screening.
* Subjects who have clinically significant cardiovascular condition.
* Subjects who have a clinically significant abnormal 12-lead ECG that results in active medical problem which may impact the safety of the patient according to Investigator's judgment.
* Subjects whose 12-lead ECG shows Fridericia's corrected QT interval (QTcF) >450 ms for males or QTcF >470 ms for females at screening or randomization visits.
* Subjects with known intolerance/hypersensitivity or contra-indication to treatment with inhaled β2-adrenergic receptor agonists, corticosteroids or propellant gases/excipients.
* Subjects with concomitant immunosuppressive therapy, use of oral or injected corticosteroids, anti- Immunoglobulin E (IgE), anti-Interleukin 5 (IL5) or other monoclonal or polyclonal antibodies within 12 weeks prior to screening.
* Use of potent cytochrome P450 3A4 inhibitors and inducers within 4 weeks prior to screening.
* History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening.
* Subjects who have received an investigational drug within 1 month or 5 half-lives (whichever is greater) prior to screening visit, or have been previously randomized in this trial, or are currently participating in another clinical trial.
* Subjects who are mentally or legally incapacitated or subjects accommodated in an establishment as a result of an official or judicial order.
* Subjects who have undergone major surgery in the 3 months prior to screening visit or have a planned surgery during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sterling, Principal Investigator — Sterling ENT, PA
Locations (10):
- United States (10):
  - Chiesi Investigational Site, Tucson, Arizona
  - Chiesi Investigational Site, Los Angeles, California
  - Chiesi Investigational Site, Lutherville, Maryland
  - Chiesi Investigational Site, St Louis, Missouri
  - Chiesi Investigational Site, Raleigh, North Carolina
  - Chiesi Investigational Site, Greenville, South Carolina
  - Chiesi Investigational Site, Orangeburg, South Carolina
  - Chiesi Investigational Site, Spartanburg, South Carolina
  - Chiesi Investigational Site, Knoxville, Tennessee
  - Chiesi Investigational Site, Richland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604
- [Background] Tilert T, Dillon C, Paulose-Ram R, Hnizdo E, Doney B. Estimating the U.S. prevalence of chronic obstructive pulmonary disease using pre- and post-bronchodilator spirometry: the National Health and Nutrition Examination Survey (NHANES) 2007-2010. Respir Res. 2013 Oct 9;14(1):103. doi: 10.1186/1465-9921-14-103. PMID 24107140
- [Background] Mannino DM. COPD: epidemiology, prevalence, morbidity and mortality, and disease heterogeneity. Chest. 2002 May;121(5 Suppl):121S-126S. doi: 10.1378/chest.121.5_suppl.121s. PMID 12010839
- [Background] Tonnesen P. Smoking cessation and COPD. Eur Respir Rev. 2013 Mar 1;22(127):37-43. doi: 10.1183/09059180.00007212. PMID 23457163
- [Background] van Eerd EA, van der Meer RM, van Schayck OC, Kotz D. Smoking cessation for people with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2016 Aug 20;2016(8):CD010744. doi: 10.1002/14651858.CD010744.pub2. PMID 27545342
- [Background] Kew KM, Mavergames C, Walters JA. Long-acting beta2-agonists for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2013 Oct 15;2013(10):CD010177. doi: 10.1002/14651858.CD010177.pub2. PMID 24127118
- [Background] McGarvey L, Niewoehner D, Magder S, Sachs P, Tetzlaff K, Hamilton A, Korducki L, Bothner U, Vogelmeier C, Koch A, Ferguson GT. One-Year Safety of Olodaterol Once Daily via Respimat(R) in Patients with GOLD 2-4 Chronic Obstructive Pulmonary Disease: Results of a Pre-Specified Pooled Analysis. COPD. 2015;12(5):484-93. doi: 10.3109/15412555.2014.991864. Epub 2015 Feb 18. PMID 25692310
- [Background] Dahl R, Chung KF, Buhl R, Magnussen H, Nonikov V, Jack D, Bleasdale P, Owen R, Higgins M, Kramer B; INVOLVE (INdacaterol: Value in COPD: Longer Term Validation of Efficacy and Safety) Study Investigators. Efficacy of a new once-daily long-acting inhaled beta2-agonist indacaterol versus twice-daily formoterol in COPD. Thorax. 2010 Jun;65(6):473-9. doi: 10.1136/thx.2009.125435. PMID 20522841
- [Background] Keating GM. Tiotropium bromide inhalation powder: a review of its use in the management of chronic obstructive pulmonary disease. Drugs. 2012 Jan 22;72(2):273-300. doi: 10.2165/11208620-000000000-00000. PMID 22217233
- [Background] Casaburi R, Kukafka D, Cooper CB, Witek TJ Jr, Kesten S. Improvement in exercise tolerance with the combination of tiotropium and pulmonary rehabilitation in patients with COPD. Chest. 2005 Mar;127(3):809-17. doi: 10.1378/chest.127.3.809. PMID 15764761
- [Background] Kesten S, Casaburi R, Kukafka D, Cooper CB. Improvement in self-reported exercise participation with the combination of tiotropium and rehabilitative exercise training in COPD patients. Int J Chron Obstruct Pulmon Dis. 2008;3(1):127-36. doi: 10.2147/copd.s2389. PMID 18488436
- [Background] Karner C, Chong J, Poole P. Tiotropium versus placebo for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD009285. doi: 10.1002/14651858.CD009285.pub2. PMID 22786525
- [Background] Wedzicha JA, Banerji D, Chapman KR, Vestbo J, Roche N, Ayers RT, Thach C, Fogel R, Patalano F, Vogelmeier CF; FLAME Investigators. Indacaterol-Glycopyrronium versus Salmeterol-Fluticasone for COPD. N Engl J Med. 2016 Jun 9;374(23):2222-34. doi: 10.1056/NEJMoa1516385. Epub 2016 May 15. PMID 27181606
- [Background] Yang IA, Clarke MS, Sim EH, Fong KM. Inhaled corticosteroids for stable chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD002991. doi: 10.1002/14651858.CD002991.pub3. PMID 22786484
- [Background] Kew KM, Seniukovich A. Inhaled steroids and risk of pneumonia for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2014 Mar 10;2014(3):CD010115. doi: 10.1002/14651858.CD010115.pub2. PMID 24615270
- [Background] Yawn BP, Li Y, Tian H, Zhang J, Arcona S, Kahler KH. Inhaled corticosteroid use in patients with chronic obstructive pulmonary disease and the risk of pneumonia: a retrospective claims data analysis. Int J Chron Obstruct Pulmon Dis. 2013;8:295-304. doi: 10.2147/COPD.S42366. Epub 2013 Jun 27. PMID 23836970
- [Background] Rachelefsky GS, Liao Y, Faruqi R. Impact of inhaled corticosteroid-induced oropharyngeal adverse events: results from a meta-analysis. Ann Allergy Asthma Immunol. 2007 Mar;98(3):225-38. doi: 10.1016/S1081-1206(10)60711-9. PMID 17378253
- [Background] Roland NJ, Bhalla RK, Earis J. The local side effects of inhaled corticosteroids: current understanding and review of the literature. Chest. 2004 Jul;126(1):213-9. doi: 10.1378/chest.126.1.213. PMID 15249465
- [Background] Tashkin DP, Murray HE, Skeans M, Murray RP. Skin manifestations of inhaled corticosteroids in COPD patients: results from Lung Health Study II. Chest. 2004 Oct;126(4):1123-33. doi: 10.1016/S0012-3692(15)31287-3. PMID 15486373
- [Background] Crim C, Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Willits LR, Yates JC, Vestbo J. Pneumonia risk in COPD patients receiving inhaled corticosteroids alone or in combination: TORCH study results. Eur Respir J. 2009 Sep;34(3):641-7. doi: 10.1183/09031936.00193908. Epub 2009 May 14. PMID 19443528
- [Background] Crim C, Dransfield MT, Bourbeau J, Jones PW, Hanania NA, Mahler DA, Vestbo J, Wachtel A, Martinez FJ, Barnhart F, Lettis S, Calverley PM. Pneumonia risk with inhaled fluticasone furoate and vilanterol compared with vilanterol alone in patients with COPD. Ann Am Thorac Soc. 2015 Jan;12(1):27-34. doi: 10.1513/AnnalsATS.201409-413OC. PMID 25490706
- [Background] Pavord ID, Lettis S, Anzueto A, Barnes N. Blood eosinophil count and pneumonia risk in patients with chronic obstructive pulmonary disease: a patient-level meta-analysis. Lancet Respir Med. 2016 Sep;4(9):731-741. doi: 10.1016/S2213-2600(16)30148-5. Epub 2016 Jul 23. PMID 27460163
- [Background] Johnell O, Pauwels R, Lofdahl CG, Laitinen LA, Postma DS, Pride NB, Ohlsson SV. Bone mineral density in patients with chronic obstructive pulmonary disease treated with budesonide Turbuhaler. Eur Respir J. 2002 Jun;19(6):1058-63. doi: 10.1183/09031936.02.00276602. PMID 12108857
- [Background] Ferguson GT, Calverley PMA, Anderson JA, Jenkins CR, Jones PW, Willits LR, Yates JC, Vestbo J, Celli B. Prevalence and progression of osteoporosis in patients with COPD: results from the TOwards a Revolution in COPD Health study. Chest. 2009 Dec;136(6):1456-1465. doi: 10.1378/chest.08-3016. Epub 2009 Jul 6. PMID 19581353
- [Background] Loke YK, Cavallazzi R, Singh S. Risk of fractures with inhaled corticosteroids in COPD: systematic review and meta-analysis of randomised controlled trials and observational studies. Thorax. 2011 Aug;66(8):699-708. doi: 10.1136/thx.2011.160028. Epub 2011 May 20. PMID 21602540
- [Background] Suissa S, Kezouh A, Ernst P. Inhaled corticosteroids and the risks of diabetes onset and progression. Am J Med. 2010 Nov;123(11):1001-6. doi: 10.1016/j.amjmed.2010.06.019. Epub 2010 Oct 1. PMID 20870201
- [Background] Wang JJ, Rochtchina E, Tan AG, Cumming RG, Leeder SR, Mitchell P. Use of inhaled and oral corticosteroids and the long-term risk of cataract. Ophthalmology. 2009 Apr;116(4):652-7. doi: 10.1016/j.ophtha.2008.12.001. Epub 2009 Feb 25. PMID 19243828
- [Background] Miller DP, Watkins SE, Sampson T, Davis KJ. Long-term use of fluticasone propionate/salmeterol fixed-dose combination and incidence of cataracts and glaucoma among chronic obstructive pulmonary disease patients in the UK General Practice Research Database. Int J Chron Obstruct Pulmon Dis. 2011;6:467-76. doi: 10.2147/COPD.S14247. Epub 2011 Sep 16. PMID 22003292
- [Background] Andrejak C, Nielsen R, Thomsen VO, Duhaut P, Sorensen HT, Thomsen RW. Chronic respiratory disease, inhaled corticosteroids and risk of non-tuberculous mycobacteriosis. Thorax. 2013 Mar;68(3):256-62. doi: 10.1136/thoraxjnl-2012-201772. Epub 2012 Jul 10. PMID 22781123
- [Background] Aaron SD, Vandemheen KL, Fergusson D, Maltais F, Bourbeau J, Goldstein R, Balter M, O'Donnell D, McIvor A, Sharma S, Bishop G, Anthony J, Cowie R, Field S, Hirsch A, Hernandez P, Rivington R, Road J, Hoffstein V, Hodder R, Marciniuk D, McCormack D, Fox G, Cox G, Prins HB, Ford G, Bleskie D, Doucette S, Mayers I, Chapman K, Zamel N, FitzGerald M; Canadian Thoracic Society/Canadian Respiratory Clinical Research Consortium. Tiotropium in combination with placebo, salmeterol, or fluticasone-salmeterol for treatment of chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):545-55. doi: 10.7326/0003-4819-146-8-200704170-00152. Epub 2007 Feb 19. PMID 17310045
- [Background] Singh D, Brooks J, Hagan G, Cahn A, O'Connor BJ. Superiority of "triple" therapy with salmeterol/fluticasone propionate and tiotropium bromide versus individual components in moderate to severe COPD. Thorax. 2008 Jul;63(7):592-8. doi: 10.1136/thx.2007.087213. Epub 2008 Feb 1. PMID 18245142
- [Background] Hanania NA, Crater GD, Morris AN, Emmett AH, O'Dell DM, Niewoehner DE. Benefits of adding fluticasone propionate/salmeterol to tiotropium in moderate to severe COPD. Respir Med. 2012 Jan;106(1):91-101. doi: 10.1016/j.rmed.2011.09.002. Epub 2011 Oct 29. PMID 22040533
- [Background] Frith PA, Thompson PJ, Ratnavadivel R, Chang CL, Bremner P, Day P, Frenzel C, Kurstjens N; Glisten Study Group. Glycopyrronium once-daily significantly improves lung function and health status when combined with salmeterol/fluticasone in patients with COPD: the GLISTEN study, a randomised controlled trial. Thorax. 2015 Jun;70(6):519-27. doi: 10.1136/thoraxjnl-2014-206670. Epub 2015 Apr 3. PMID 25841237
- [Background] Siler TM, Kerwin E, Singletary K, Brooks J, Church A. Efficacy and Safety of Umeclidinium Added to Fluticasone Propionate/Salmeterol in Patients with COPD: Results of Two Randomized, Double-Blind Studies. COPD. 2016;13(1):1-10. doi: 10.3109/15412555.2015.1034256. Epub 2015 Oct 9. PMID 26451734
- [Background] Singh D, Papi A, Corradi M, Pavlisova I, Montagna I, Francisco C, Cohuet G, Vezzoli S, Scuri M, Vestbo J. Single inhaler triple therapy versus inhaled corticosteroid plus long-acting beta2-agonist therapy for chronic obstructive pulmonary disease (TRILOGY): a double-blind, parallel group, randomised controlled trial. Lancet. 2016 Sep 3;388(10048):963-73. doi: 10.1016/S0140-6736(16)31354-X. Epub 2016 Sep 1. PMID 27598678
- [Background] Nelson HS, Weiss ST, Bleecker ER, Yancey SW, Dorinsky PM; SMART Study Group. The Salmeterol Multicenter Asthma Research Trial: a comparison of usual pharmacotherapy for asthma or usual pharmacotherapy plus salmeterol. Chest. 2006 Jan;129(1):15-26. doi: 10.1378/chest.129.1.15. PMID 16424409
- [Background] Wijesinghe M, Weatherall M, Perrin K, Harwood M, Beasley R. Risk of mortality associated with formoterol: a systematic review and meta-analysis. Eur Respir J. 2009 Oct;34(4):803-11. doi: 10.1183/09031936.00159708. PMID 19797669
- [Background] Chowdhury BA, Dal Pan G. The FDA and safe use of long-acting beta-agonists in the treatment of asthma. N Engl J Med. 2010 Apr 1;362(13):1169-71. doi: 10.1056/NEJMp1002074. Epub 2010 Feb 24. No abstract available. PMID 20181964
- [Background] Drazen JM, O'Byrne PM. Risks of long-acting beta-agonists in achieving asthma control. N Engl J Med. 2009 Apr 16;360(16):1671-2. doi: 10.1056/NEJMe0902057. No abstract available. PMID 19369675
- [Background] Chowdhury BA, Seymour SM, Levenson MS. Assessing the safety of adding LABAs to inhaled corticosteroids for treating asthma. N Engl J Med. 2011 Jun 30;364(26):2473-5. doi: 10.1056/NEJMp1104375. No abstract available. PMID 21714647
- [Background] Stempel DA, Raphiou IH, Kral KM, Yeakey AM, Emmett AH, Prazma CM, Buaron KS, Pascoe SJ; AUSTRI Investigators. Serious Asthma Events with Fluticasone plus Salmeterol versus Fluticasone Alone. N Engl J Med. 2016 May 12;374(19):1822-30. doi: 10.1056/NEJMoa1511049. Epub 2016 Mar 6. PMID 26949137
- [Background] Stempel DA, Szefler SJ, Pedersen S, Zeiger RS, Yeakey AM, Lee LA, Liu AH, Mitchell H, Kral KM, Raphiou IH, Prillaman BA, Buaron KS, Yun Kirby S, Pascoe SJ; VESTRI Investigators. Safety of Adding Salmeterol to Fluticasone Propionate in Children with Asthma. N Engl J Med. 2016 Sep 1;375(9):840-9. doi: 10.1056/NEJMoa1606356. PMID 27579634
- [Background] Novartis Pharma. FORADIL®AEROLIZER® US Prescribing Information. Whitehouse Station, New Jersey; 2012 Sep.
- [Background] Chiesi Farmaceutici S.p.A. A randomized, double blind, double dummy, cumulative dose, safety cross-over trial comparing 4 increasing doses of Formoterol-HFA (pMDI) versus 4 increasing doses of formoterol-DPI (Aerolizer®) and placebo (pMDI or Aerolizer ®) in asthmatic patients. RA/PR/3301/002/01.
- [Background] Chiesi Farmaceutici S.p.A. A randomized, double blind, double dummy, single dose, crossover trial comparing the efficacy and safety of a single dose administered via 1 puff of 6 μg or 2 puffs of 6 μg of formoterol-HFA (pMDI) versus a single dose of 12 μg of formoterol- DPI (Foradil®Aerolizer®) and of placebo (pMDI or Aerolizer®) in moderate to severe asthmatic patients. RA/PR/3301/009/03.
- [Background] Bensch G, Lapidus RJ, Levine BE, Lumry W, Yegen U, Kiselev P, Della Cioppa G. A randomized, 12-week, double-blind, placebo-controlled study comparing formoterol dry powder inhaler with albuterol metered-dose inhaler. Ann Allergy Asthma Immunol. 2001 Jan;86(1):19-27. doi: 10.1016/s1081-1206(10)62351-4. PMID 11206232
- [Background] Pleskow W, LaForce CF, Yegen U, Matos D, Della Cioppa G. Formoterol delivered via the dry powder Aerolizer inhaler versus albuterol MDI and placebo in mild-to-moderate asthma: a randomized, double-blind, double-dummy trial. J Asthma. 2003;40(5):505-14. doi: 10.1081/jas-120018780. PMID 14529100
- [Background] Dahl R, Greefhorst LA, Nowak D, Nonikov V, Byrne AM, Thomson MH, Till D, Della Cioppa G; Formoterol in Chronic Obstructive Pulmonary Disease I Study Group. Inhaled formoterol dry powder versus ipratropium bromide in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Sep 1;164(5):778-84. doi: 10.1164/ajrccm.164.5.2007006. PMID 11549532
- [Background] Rossi A, Kristufek P, Levine BE, Thomson MH, Till D, Kottakis J, Della Cioppa G; Formoterol in Chronic Obstructive Pulmonary Disease (FICOPD) II Study Group. Comparison of the efficacy, tolerability, and safety of formoterol dry powder and oral, slow-release theophylline in the treatment of COPD. Chest. 2002 Apr;121(4):1058-69. doi: 10.1378/chest.121.4.1058. PMID 11948033
- [Background] Mylan Specialty L.P. PERFOROMIST® US Prescribing Information. Morgantown, West Virginia; 2013 Mar.
- [Background] Gross NJ, Nelson HS, Lapidus RJ, Dunn L, Lynn L, Rinehart M, Denis-Mize K; Formoterol Study Group. Efficacy and safety of formoterol fumarate delivered by nebulization to COPD patients. Respir Med. 2008 Feb;102(2):189-97. doi: 10.1016/j.rmed.2007.10.007. PMID 18363201
- [Background] Chiesi Farmaceutici S.p.A. CHF 1535 HFA : BDP + formoterol 100/6 μg pressurized inhalation solution : Common Technical Document. Module 2.5: 8.
- [Background] Bousquet J, Guenole E, Duvauchelle T, Vicaut E, Lefrancois G. A randomized, double-blind, double-dummy, single-dose, crossover trial evaluating the efficacy and safety profiles of two dose levels (12 and 24 microg) of formoterol-HFA (pMDI) vs. those of a dose level (24 microg) of formoterol-DPI (Foradil/Aerolizer) and of placebo (pMDI or Aerolizer) in moderate to severe asthmatic patients. Respiration. 2005;72 Suppl 1:13-9. doi: 10.1159/000083688. PMID 15915008
- [Background] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Background] Houghton CM, Langley SJ, Singh SD, Holden J, Monici Preti AP, Acerbi D, Poli G, Woodcock A. Comparison of bronchoprotective and bronchodilator effects of a single dose of formoterol delivered by hydrofluoroalkane and chlorofluorocarbon aerosols and dry powder in a double blind, placebo-controlled, crossover study. Br J Clin Pharmacol. 2004 Oct;58(4):359-66. doi: 10.1111/j.1365-2125.2004.02172.x. PMID 15373928
- [Background] Juniper EF, Bousquet J, Abetz L, Bateman ED; GOAL Committee. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. Respir Med. 2006 Apr;100(4):616-21. doi: 10.1016/j.rmed.2005.08.012. Epub 2005 Oct 13. PMID 16226443
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Arievich H, Overend T, Renard D, Gibbs M, Alagappan V, Looby M, Banerji D. A novel model-based approach for dose determination of glycopyrronium bromide in COPD. BMC Pulm Med. 2012 Dec 8;12:74. doi: 10.1186/1471-2466-12-74. PMID 23217058
- [Background] Center for Drug Evaluation and Research Medical Review. Clinical Team Leader Memorandum: Formoterol fumarate inhalation solution 20mcg/2mL; NDA # 22-007: 2007 Mar 15.
- [Background] Gross NJ, Kerwin E, Levine B, Kim KT, Denis-Mize K, Hamzavi M, Carpenter M, Rinehart M. Nebulized formoterol fumarate: Dose selection and pharmacokinetics. Pulm Pharmacol Ther. 2008 Oct;21(5):818-23. doi: 10.1016/j.pupt.2008.07.002. Epub 2008 Jul 8. PMID 18655841
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Hankinson JL, Kawut SM, Shahar E, Smith LJ, Stukovsky KH, Barr RG. Performance of American Thoracic Society-recommended spirometry reference values in a multiethnic sample of adults: the multi-ethnic study of atherosclerosis (MESA) lung study. Chest. 2010 Jan;137(1):138-45. doi: 10.1378/chest.09-0919. Epub 2009 Sep 9. PMID 19741060
- [Background] Hankinson JL, Bang KM. Acceptability and reproducibility criteria of the American Thoracic Society as observed in a sample of the general population. Am Rev Respir Dis. 1991 Mar;143(3):516-21. doi: 10.1164/ajrccm/143.3.516. PMID 2001060
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] Virchow JC, Backer V, de Blay F, Kuna P, Ljorring C, Prieto JL, Villesen HH. Defining moderate asthma exacerbations in clinical trials based on ATS/ERS joint statement. Respir Med. 2015 May;109(5):547-56. doi: 10.1016/j.rmed.2015.01.012. Epub 2015 Feb 3. PMID 25676887
- [Background] Edwards D, Berry JJ. The efficiency of simulation-based multiple comparisons. Biometrics. 1987 Dec;43(4):913-28. PMID 3427176
- See also: Global Initiative for Chronic Obstructive Lung Disease, Inc. Global strategy for the diagnosis, management, and prevention of Chronic Obstructive Pulmonary Disease: 2017 — http://goldcopd.org/
- See also: Global Initiative for Asthma. Global strategy for asthma management and prevention (2016 update). 2016. — http://www.ginasthma.org
- See also: Centers for Disease Control and Prevention: Asthma — https://www.cdc.gov/asthma/most_recent_data.htm
- See also: Chiesi Farmaceutici S.p.A Respiratory — https://www.chiesi.com/en/air/
- See also: Chiesi Farmaceutici S.p.A - Press Release: Chiesi Farmaceutifici is the first company to submit a marketing authorisation application to the European Medicine Agency for a triple combination for the treatment of COPD — https://www.chiesi.com/en/chiesi-farmaceutici-is-the-first-company-to-submit-a-marketing-authorisation-application-to-the-european-medicine-agency-for-a-triple-combination-for-the-treatment-of-copd-
- See also: RT Magazine: Asthma-COPD Therapy Foradil Aerolizer to be Discontinued — http://www.rtmagazine.com/2015/10/asthma-copd-foradil-aerolizer-to-be-discontinued/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with confirmed diagnosis of asthma were recruited into the study according to the trial inclusion and exclusion criteria and were randomized into one of the 6 treatment groups. The total daily dose (TDD) of the trial investigational drug CHF 1531 pressurized metered dose Inhaler (pMDI), inhalation solution (IS) of the direct comparator, or matched placebo is indicated for each treatment group.
Groups:
- Overall Study Group: Each eligible patient was randomly assigned to one of the 12 treatments sequences. The study had an incomplete cross-over design. Patients were planned to take 4 out of 6 treatments, according to one of 12 possible sequences using a balanced incomplete block randomization scheme. Treatment intervals were separated by 2-week wash-out periods.
  For clarity, a summary of study participants who received treatment A, B, C, D, E, and F is presented below as milestones and also as periods.
Period: Study Participants
Arm/Group | Overall Study Group
Started (Due to an error in the randomization system during the trial, some patients received the same treatment in several treatment intervals. The error was recognized after the database lock and unblinding. Patients were analyzed according to the treatments assigned by the Interactive Response Technology (IRT) system. For statistical analyses "as randomized" corresponds to "as actually allocated by the IRT" that was used for efficacy analyses not according to those which were originally planned.) | 67
Treatment A (Number of patients who received Treatment A.) | 39
Treatment B (Number of patients who received Treatment B.) | 35
Treatment C (Number of patients who received Treatment C.) | 37
Treatment D (Number of patients who received Treatment D.) | 40
Treatment E (Number of patients who received Treatment E.) | 40
Treatment F (Number of patients who received Treatment F.) | 41
Completed (Patients who received the same treatment during two treatment intervals were considered twice in the corresponding group (once for each treatment interval). The table above presents the number of patients receiving each treatment in at least one treatment interval.) | 58
Not Completed | 9
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 6
Period: Treatment A
Arm/Group | Overall Study Group
Started | 39
Completed | 35
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Period: Treatment B
Arm/Group | Overall Study Group
Started | 35
Completed | 35
Not Completed | 0
Period: Treatment C
Arm/Group | Overall Study Group
Started | 37
Completed | 35
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Treatment D
Arm/Group | Overall Study Group
Started | 40
Completed | 40
Not Completed | 0
Period: Treatment E
Arm/Group | Overall Study Group
Started | 40
Completed | 36
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Period: Treatment F
Arm/Group | Overall Study Group
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT): All randomized patients who received at least one dose of the study treatment within the given period and with at least one available evaluation of efficacy (primary or secondary efficacy variables) after the baseline and within the given period.
Groups:
- Trial Participants: All trial participants had diagnosed asthma and were randomized to 6 treatments in a cross-over study design.
Arm/Group | Trial Participants
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 67
Weight [Mean (Standard Deviation); unit: kg] | 89.8 (23.1)
Height [Mean (Standard Deviation); unit: cm] | 167.6 (10.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.0 (8.1)
Time since first diagnosis of asthma [Median (Full Range); unit: months] | 335.2 [80.8 to 810.4]
Age at first diagnosis of asthma [Mean (Standard Deviation); unit: years] | 17.3 (17.4)
Asthma medication category at study entry [Count of Participants; unit: Participants]
  Short-acting beta2-agonist (SABA [albuterol]) | 62
  Leukotriene modifiers (LTRM) | 7
  Theophylline | 0
  Inhaled corticosteroid (ICS) alone | 27
  ICS/Long-acting muscarinic antagonist (LABA), (free or fixed combination) | 39
  ICS/Long-acting muscarinic antagonist (LAMA), (free combination) | 1
  ICS/LABA/LAMA | 0
Smoking habits [Count of Participants; unit: Participants]
  Current smoker | 0
  Ex-smoker | 9
  Non-smoker | 58
Duration of smoking [Mean (Standard Deviation); unit: years] — Population: Only 9 trial participants had smoked (ex-smokers); thus, results on 9 participants are reported.
  years
    number analyzed (Participants) | 9
    (all) | 8.0 (4.5)
Number of pack-years [Median (Full Range); unit: pack-years] — Population: Only 9 trial participants had smoked (ex-smokers).
  pack-years
    number analyzed (Participants) | 9
    (all) | 2.5 [0.5 to 9.0]
FEV1 at screening (pre-bronchodilator) [Mean (Standard Deviation); unit: Litre] — Measure description: Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath during the first second (i.e. FEV1) of the expiratory maneuver.
  Litre | 2.128 (0.620)
FEV1 % of the normal predicted value (pre-bronchodilator) [Mean (Standard Deviation); unit: percent] | 70.2 (6.3)
FEV1 at screening (post-bronchodilator) [Mean (Standard Deviation); unit: Litre] | 2.548 (0.738)
FEV1 % of the normal predicted value (post-bronchodilator) [Mean (Standard Deviation); unit: percent] | 84.2 (8.1)
FVC at screening (pre-bronchodilator) [Mean (Standard Deviation); unit: Litre] — Measure description: Forced vital capacity (FVC) is the maximal volume of gas that can be exhaled from full inhalation by exhaling as forcefully and rapidly as possible.
  Litre | 3.066 (0.993)
FVC at screening (post-bronchodilator) [Mean (Standard Deviation); unit: Litre] | 3.450 (1.028)
Reversibility FEV1 (mL) at screening [Mean (Standard Deviation); unit: millilitre] | 420 (178)
Reversibility FEV1 (%) at screening [Mean (Standard Deviation); unit: percent] | 20.1 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Area Under the Curve Between 0 and 12 h [AUC(0-12h)], Normalized by Time -- Change From Baseline to Post Dose Day 14
Description: Spirometry used to measure FEV1, was performed according to internationally accepted standards. Results show the change from baseline in FEV1 AUC(0-12h), normalized by time on Day 14; it was calculated by using the linear trapezoidal rule, based on the changes in FEV1 from the baseline values.
  Patients receiving the same treatment during two periods are considered twice in the ANCOVA model (once for each period attended).
  Definitions:
  AUC=Area under the curve; AUC(0-12h)=AUC between 0 and 12 h; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose) on Day 1 of the treatment period; FEV1=Forced expiratory volume in the 1st second;
Time Frame: Baseline, Day 14 post-dose
Population: Intention-to-treat (ITT): All randomized patients who received at least one dose of the study treatment within the given treatment period and with at least one available evaluation of efficacy (primary or secondary efficacy variables) after the baseline and within the given treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Groups:
- Treatment A: Treatment A, CHF 1531 pMDI: 6 μg TDD
- Treatment B: Treatment B, CHF 1531 pMDI: 12 μg TDD
- Treatment C: Treatment C, CHF 1531 pMDI: 24 μg TDD
- Treatment D: Treatment D, CHF 1531 pMDI: 48 μg TDD
- Treatment E: Treatment E, Matched placebo
- Treatment F: Treatment F, Formoterol fumarate IS Perforomist®: 40 μg TDD
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
Litres | 0.174 [0.141 to 0.208] | 0.221 [0.186 to 0.257] | 0.197 [0.161 to 0.232] | 0.231 [0.199 to 0.263] | 0.064 [0.030 to 0.098] | 0.208 [0.175 to 0.240]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Comparison groups were: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). The primary endpoint was analyzed using an analysis of covariance (ANCOVA) including treatment, period, and patient as fixed effects and baseline as a covariate. The confidence intervals (CIs) and the p-values of the comparisons between each dose of CHF 1531 pMDI and Placebo at Day 14 were adjusted for multiplicity, based on the parametric simulation method of Edwards and Berry; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [0.050 to 0.171]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.158, 95% CI 2-sided [0.095 to 0.220]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.133, 95% CI 2-sided [0.072 to 0.194]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.167, 95% CI 2-sided [0.109 to 0.225]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison groups were: Treatment F ( Perforomist® IS 40 μg TDD) versus Treatment E (Placebo). The statistical analysis was performed using an analysis of covariance (ANCOVA) including treatment, period, and patient as fixed effects, and baseline as a covariate; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [0.098 to 0.190]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). The statistical analysis was performed using an analysis of covariance (ANCOVA) including treatment, period, and patient as fixed effects, and baseline as a covariate; Test type: Superiority; p = 0.059, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [-0.002 to 0.095]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #6 of this outcome measure; Test type: Superiority; p = 0.361, ANCOVA; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.026 to 0.070]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #6 of this outcome measure; Test type: Superiority; p = 0.016, ANCOVA; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [0.011 to 0.102]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #6 of this outcome measure; Test type: Superiority; p = 0.340, ANCOVA; Mean Difference (Final Values) = -0.025, 95% CI 2-sided [-0.075 to 0.026]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #6 of this outcome measure; Test type: Superiority; p = 0.690, ANCOVA; Mean Difference (Final Values) = 0.010, 95% CI 2-sided [-0.038 to 0.058]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment C (CHF 1531 pMDI 24 μg TDD). Statistical analysis was performed as described for the statistical analysis #6 of this outcome measure; Test type: Superiority; p = 0.155, ANCOVA; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.013 to 0.082]

2. Primary Outcome: Sensitivity Analysis 1: FEV1 AUC(0-12h), Normalized by Time -- Change From Baseline to Post Dose Day 14
Description: The primary analysis was repeated, considering patients "as randomized" and including only the first instance of each treatment.
  Patients receiving the same treatment in more than one period were included in the analysis with only data from the first instance of each treatment.
Time Frame: Baseline, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
Litres | 0.169 [0.134 to 0.205] | 0.224 [0.187 to 0.260] | 0.196 [0.158 to 0.233] | 0.232 [0.198 to 0.265] | 0.058 [0.021 to 0.094] | 0.206 [0.173 to 0.239]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Comparison groups: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). Analysis of covariance model: treatment, subject, and period as fixed effects; baseline FEV1 value as covariates. CIs and p-values for CHF 1531 pMDI vs Placebo are adjusted for multiplicity (parametric simulation method by Edwards and Berry). Subjects receiving the same treatment in more than one period are included in the primary efficacy model with only data from the first instance of each treatment; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [0.049 to 0.175]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.166, 95% CI 2-sided [0.101 to 0.230]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.138, 95% CI 2-sided [0.074 to 0.203]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [0.113 to 0.235]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison groups were: Treatment F ( Perforomist® IS 40 μg TDD) versus Treatment E (Placebo). Analysis of covariance model: treatment, subject, and period as fixed effects; baseline FEV1 value as covariates. Subjects receiving the same treatment in more than one period are included in the primary efficacy model with only data from the first instance of each treatment; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.149, 95% CI 2-sided [0.101 to 0.197]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Analysis of covariance model: treatment, subject, and period as fixed effects; baseline FEV1 value as covariates. Subjects receiving the same treatment in more than one period are included in the primary efficacy model with only data from the first instance of each treatment; Test type: Superiority; p = 0.035, ANCOVA; Mean Difference (Final Values) = 0.054, 95% CI 2-sided [0.004 to 0.104]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.301, ANCOVA; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.024 to 0.076]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Final Values) = 0.062, 95% CI 2-sided [0.014 to 0.110]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.294, ANCOVA; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.080 to 0.024]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.747, ANCOVA; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.042 to 0.058]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 11]; Test type: Superiority; p = 0.155, ANCOVA; Mean Difference (Final Values) = 0.036, 95% CI 2-sided [-0.014 to 0.086]

3. Primary Outcome: Sensitivity Analysis 2: FEV1 AUC(0-12h), Normalized by Time -- Change From Baseline to Post Dose Day 14
Description: The primary analysis was repeated, considering only patients and treatment periods for which treatment was assigned on or after the randomization error occurred.
  The number of patients shown represents those with at least one post-baseline assessment available.
Time Frame: Baseline, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 31 | 27 | 28 | 34 | 32 | 30
Litres | 0.129 [0.089 to 0.170] | 0.180 [0.136 to 0.223] | 0.159 [0.116 to 0.201] | 0.179 [0.141 to 0.217] | -0.006 [-0.047 to 0.034] | 0.170 [0.129 to 0.211]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). Analysis of covariance model: treatment, subject, and period as fixed effects; baseline FEV1 value as covariates. CIs and p-values for CHF 1531 pMDI vs Placebo are adjusted for multiplicity (parametric simulation method by Edwards and Berry). Subjects receiving the same treatment in more than one period are included in the model with only data for the instance of each treatment, which occurred after the randomization error; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.136, 95% CI 2-sided [0.065 to 0.207]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.186, 95% CI 2-sided [0.113 to 0.258]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.165, 95% CI 2-sided [0.092 to 0.238]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.185, 95% CI 2-sided [0.118 to 0.252]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison groups were: Treatment F ( Perforomist® IS 40 μg TDD) versus Treatment E (Placebo). Analysis of covariance model: treatment, subject, and period as fixed effects; baseline FEV1 value as covariates. Subjects receiving the same treatment in more than one period are included in the model with only data for the instance of each treatment which occurred after the randomization error; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.176, 95% CI 2-sided [0.121 to 0.231]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Analysis of covariance model: treatment, subject, and period as fixed effects; baseline FEV1 value as covariates. Subjects receiving the same treatment in more than one period are included in the model with only data for the instance of each treatment which occurred after the randomization error; Test type: Superiority; p = 0.088, ANCOVA; Mean Difference (Final Values) = 0.050, 95% CI 2-sided [-0.008 to 0.108]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.323, ANCOVA; Mean Difference (Final Values) = 0.029, 95% CI 2-sided [-0.029 to 0.088]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.073, ANCOVA; Mean Difference (Final Values) = 0.049, 95% CI 2-sided [-0.005 to 0.103]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.489, ANCOVA; Mean Difference (Final Values) = -0.021, 95% CI 2-sided [-0.080 to 0.039]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.978, ANCOVA; Median Difference (Final Values) = -0.001, 95% CI 2-sided [-0.057 to 0.056]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 11]; Test type: Superiority; p = 0.484, ANCOVA; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.037 to 0.077]

4. Primary Outcome: Sensitivity Analysis 3: FEV1 AUC(0-12h), Normalized by Time -- Change From Baseline to Post Dose Day 14
Description: Patients receiving the same treatment during two treatment periods are considered twice in the ANCOVA model (once for each period attended).
  Patients considered in this analysis are those with at least one available post-baseline assessment.
Time Frame: Baseline, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
Litres | 0.144 [0.103 to 0.186] | 0.194 [0.151 to 0.237] | 0.170 [0.128 to 0.213] | 0.198 [0.157 to 0.238] | 0.037 [-0.004 to 0.079] | 0.184 [0.143 to 0.225]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Comparison groups: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). Analysis of covariance model: treatment and period as fixed effects, subject as random effect, baseline FEV1 value as covariate. CIs and p-values for CHF 1531 pMDI vs Placebo are adjusted for multiplicity (parametric simulation method by Edwards and Berry). Patients receiving the same treatment during two periods are considered twice in the ANCOVA model (once for each period attended); Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.107, 95% CI 2-sided [0.048 to 0.166]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.157, 95% CI 2-sided [0.096 to 0.217]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.133, 95% CI 2-sided [0.073 to 0.193]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.160, 95% CI 2-sided [0.103 to 0.217]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison groups were: Treatment F ( Perforomist® IS 40 μg TDD) versus Treatment E (Placebo). Analysis of covariance model: treatment and period as fixed effects, subject as random effect, baseline FEV1 value as covariate. Patients receiving the same treatment during two periods are considered twice in the ANCOVA model (once for each period attended); Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.147, 95% CI 2-sided [0.102 to 0.192]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Analysis of covariance model: treatment and period as fixed effects, subject as random effect, baseline FEV1 value as covariate. Patients receiving the same treatment during two periods are considered twice in the ANCOVA model (once for each period attended); Test type: Superiority; p = 0.041, ANCOVA; Mean Difference (Final Values) = 0.050, 95% CI 2-sided [0.002 to 0.098]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.275, ANCOVA; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.021 to 0.073]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.021, ANCOVA; Mean Difference (Final Values) = 0.053, 95% CI 2-sided [0.008 to 0.098]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 1, analysis 9]; Test type: Superiority; p = 0.350, ANCOVA; Mean Difference (Final Values) = -0.024, 95% CI 2-sided [-0.073 to 0.026]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 1, analysis 10]; Test type: Superiority; p = 0.886, ANCOVA; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.044 to 0.051]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 11]; Test type: Superiority; p = 0.254, ANCOVA; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [-0.020 to 0.074]

5. Secondary Outcome: FEV1 AUC(0-12h), Normalized by Time -- Change From Baseline to Post Dose Day 1
Description: Spirometry used to measure FEV1, was performed according to internationally accepted standards.
  Patients receiving the same treatment during two periods are considered twice in the ANCOVA model (once for each period attended).
  Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose) on Day 1 of the treatment period;
Time Frame: Baseline, Day 1 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 34 | 37 | 40 | 40 | 39
Litres | 0.181 [0.143 to 0.219] | 0.221 [0.179 to 0.262] | 0.260 [0.221 to 0.298] | 0.282 [0.245 to 0.319] | 0.067 [0.030 to 0.103] | 0.239 [0.201 to 0.277]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Comparison groups were: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). This secondary efficacy variable was analyzed using the ANCOVA model that was also used for the primary efficacy analysis, without adjusting for multiplicity; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [0.060 to 0.169]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.154, 95% CI 2-sided [0.099 to 0.208]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.193, 95% CI 2-sided [0.138 to 0.247]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.216, 95% CI 2-sided [0.163 to 0.268]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Comparison groups were: Treatment F ( Perforomist® IS 40 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.172, 95% CI 2-sided [0.120 to 0.224]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.165, ANCOVA; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.016 to 0.095]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [0.024 to 0.132]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.049 to 0.153]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.187, ANCOVA; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.019 to 0.097]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.028, ANCOVA; Mean Difference (Final Values) = 0.062, 95% CI 2-sided [0.007 to 0.116]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment C (CHF 1531 pMDI 24 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.406, ANCOVA; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.031 to 0.076]

6. Secondary Outcome: FEV1 AUC(0-4h), Normalized by Time -- Change From Baseline to Post Dose Day 1 and Day 14
Description: as for outcome 5
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Intention-to-treat (ITT): All randomized patients who received at least one dose of the study treatment within the given treatment period and with at least one available evaluation of efficacy (primary or secondary efficacy variables) after the baseline and within the given treatment period.
  Due to an error in the randomization system during the trial, some patients received the same treatment in several treatment period, as summarized in section Participant Flow.
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
Litres
  Day 1: number analyzed (Participants) | 39 | 34 | 37 | 40 | 40 | 40
  Day 1 | 0.220 [0.180 to 0.260] | 0.250 [0.207 to 0.293] | 0.270 [0.229 to 0.311] | 0.317 [0.279 to 0.356] | 0.047 [0.009 to 0.085] | 0.288 [0.249 to 0.328]
  Day 14: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14 | 0.214 [0.174 to 0.254] | 0.251 [0.210 to 0.293] | 0.231 [0.190 to 0.273] | 0.278 [0.241 to 0.316] | 0.061 [0.021 to 0.101] | 0.259 [0.221 to 0.298]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Day 1 Comparison groups were: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). This secondary efficacy variable was analyzed using the ANCOVA model that was also used for the primary efficacy analysis, without adjusting for multiplicity; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.173, 95% CI 2-sided [0.116 to 0.230]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; Day 1 Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.203, 95% CI 2-sided [0.146 to 0.260]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; Day 1 Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.223, 95% CI 2-sided [0.166 to 0.280]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; Day 1 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.270, 95% CI 2-sided [0.216 to 0.325]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; Day 1 Comparison groups were: Treatment F ( Perforomist® IS 40 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.241, 95% CI 2-sided [0.187 to 0.295]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; Day 1 Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.308, ANCOVA; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.028 to 0.089]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Day 1 Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.082, ANCOVA; Mean Difference (Final Values) = 0.050, 95% CI 2-sided [-0.006 to 0.107]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; Day 1 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.097, 95% CI 2-sided [0.043 to 0.152]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; Day 1 Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.520, ANCOVA; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.041 to 0.080]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; Day 1 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.022, ANCOVA; Mean Difference (Final Values) = 0.067, 95% CI 2-sided [0.010 to 0.124]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Day 1 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment C (CHF 1531 pMDI 24 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.098, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [-0.009 to 0.103]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; Day 14 Comparison groups were: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.153, 95% CI 2-sided [0.095 to 0.210]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; Day 14 Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.190, 95% CI 2-sided [0.131 to 0.249]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; Day 14 Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.170, 95% CI 2-sided [0.113 to 0.228]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; Day 14 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.217, 95% CI 2-sided [0.162 to 0.272]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; Day 14 Comparison groups were: Treatment F ( Perforomist® IS 40 μg TDD) versus Treatment E (Placebo). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.198, 95% CI 2-sided [0.144 to 0.252]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; Day 14 Comparison groups were: Treatment B (CHF 1531 pMDI 12 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.203, ANCOVA; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [-0.020 to 0.095]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; Day 14 Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.542, ANCOVA; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.039 to 0.074]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; Day 14 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment A (CHF 1531 pMDI 6 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.021, ANCOVA; Mean Difference (Final Values) = 0.064, 95% CI 2-sided [0.010 to 0.119]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; Day 14 Comparison groups were: Treatment C (CHF 1531 pMDI 24 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.510, ANCOVA; Mean Difference (Final Values) = -0.020, 95% CI 2-sided [-0.080 to 0.040]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; Day 14 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment B (CHF 1531 pMDI 12 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.352, ANCOVA; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [-0.030 to 0.084]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; Day 14 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment C (CHF 1531 pMDI 24 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; Test type: Superiority; p = 0.098, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [-0.009 to 0.103]

7. Secondary Outcome: FEV1 Peak(0-4h), Normalized by Time -- Change From Baseline to Post Dose Day 1 and Day 14
Description: Spirometry, used to measure FEV1, was performed according to internationally accepted standards.
  Patients receiving the same treatment during two periods are considered twice in the ANCOVA model (once for each period attended).
  Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose) on Day 1 of the treatment period;
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
Litres
  Day 1 | 0.359 [0.317 to 0.401] | 0.370 [0.326 to 0.414] | 0.393 [0.351 to 0.436] | 0.430 [0.390 to 0.470] | 0.178 [0.138 to 0.218] | 0.416 [0.375 to 0.457]
  Day 14: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14 | 0.346 [0.303 to 0.390] | 0.373 [0.328 to 0.419] | 0.349 [0.304 to 0.394] | 0.389 [0.348 to 0.430] | 0.183 [0.140 to 0.227] | 0.367 [0.325 to 0.409]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.181, 95% CI 2-sided [0.122 to 0.241]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.192, 95% CI 2-sided [0.133 to 0.251]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.215, 95% CI 2-sided [0.156 to 0.275]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.252, 95% CI 2-sided [0.195 to 0.309]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.238, 95% CI 2-sided [0.182 to 0.295]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.723, ANCOVA; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.049 to 0.071]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p = 0.257, ANCOVA; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.025 to 0.093]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.016, ANCOVA; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [0.014 to 0.128]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.464, ANCOVA; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.039 to 0.086]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.048, ANCOVA; Mean Difference (Final Values) = 0.060, 95% CI 2-sided [0.000 to 0.120]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 11]; Test type: Superiority; p = 0.219, ANCOVA; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [-0.022 to 0.095]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 12]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.163, 95% CI 2-sided [0.100 to 0.226]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.190, 95% CI 2-sided [0.126 to 0.254]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 14]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.166, 95% CI 2-sided [0.103 to 0.229]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.206, 95% CI 2-sided [0.146 to 0.266]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 16]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.184, 95% CI 2-sided [0.125 to 0.243]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.400, ANCOVA; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [-0.036 to 0.090]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 18]; Test type: Superiority; p = 0.931, ANCOVA; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.059 to 0.064]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 19]; Test type: Superiority; p = 0.160, ANCOVA; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [-0.017 to 0.102]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 20]; Test type: Superiority; p = 0.464, ANCOVA; Mean Difference (Final Values) = -0.024, 95% CI 2-sided [-0.090 to 0.041]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.623, ANCOVA; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.047 to 0.078]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.197, ANCOVA; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.021 to 0.101]

8. Secondary Outcome: FVC AUC(0-12h), Normalized by Time -- Change From Baseline to Post Dose Day 1 and Day 14
Description: Spirometry, used to measure FVC, was performed according to internationally accepted standards.
  Patients receiving the same treatment during two periods are considered twice in the ANCOVA model (once for each period attended).
  Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose) on Day 1 of the treatment period;
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
Litres
  Day 1: number analyzed (Participants) | 39 | 34 | 37 | 40 | 40 | 39
  Day 1 | 0.111 [0.068 to 0.154] | 0.156 [0.109 to 0.203] | 0.160 [0.116 to 0.204] | 0.182 [0.140 to 0.224] | 0.059 [0.018 to 0.100] | 0.172 [0.128 to 0.215]
  Day 14: number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
  Day 14 | 0.103 [0.064 to 0.142] | 0.134 [0.093 to 0.174] | 0.120 [0.079 to 0.160] | 0.142 [0.105 to 0.178] | 0.060 [0.020 to 0.099] | 0.134 [0.096 to 0.171]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.098, ANCOVA; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.010 to 0.113]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = 0.097, 95% CI 2-sided [0.035 to 0.159]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.039 to 0.163]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.122, 95% CI 2-sided [0.063 to 0.182]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [0.054 to 0.171]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.162, ANCOVA; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [-0.018 to 0.108]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p = 0.117, ANCOVA; Mean Difference (Final Values) = 0.049, 95% CI 2-sided [-0.012 to 0.110]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.020, ANCOVA; Mean Difference (Final Values) = 0.071, 95% CI 2-sided [0.011 to 0.130]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.909, ANCOVA; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.062 to 0.070]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.419, ANCOVA; Mean Difference (Final Values) = 0.025, 95% CI 2-sided [-0.037 to 0.088]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 11]; Test type: Superiority; p = 0.483, ANCOVA; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.039 to 0.083]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 12]; Test type: Superiority; p = 0.126, ANCOVA; Mean Difference (Final Values) = 0.043, 95% CI 2-sided [-0.012 to 0.099]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p = 0.012, ANCOVA; Mean Difference (Final Values) = 0.074, 95% CI 2-sided [0.017 to 0.131]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 14]; Test type: Superiority; p = 0.037, ANCOVA; Mean Difference (Final Values) = 0.060, 95% CI 2-sided [0.004 to 0.116]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [0.028 to 0.136]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 16]; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Final Values) = 0.074, 95% CI 2-sided [0.021 to 0.127]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.282, ANCOVA; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.025 to 0.087]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 18]; Test type: Superiority; p = 0.554, ANCOVA; Mean Difference (Final Values) = 0.017, 95% CI 2-sided [-0.039 to 0.072]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 19]; Test type: Superiority; p = 0.149, ANCOVA; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.014 to 0.091]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 20]; Test type: Superiority; p = 0.636, ANCOVA; Mean Difference (Final Values) = -0.014, 95% CI 2-sided [-0.072 to 0.044]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.775, ANCOVA; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.047 to 0.063]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.425, ANCOVA; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.032 to 0.077]

9. Secondary Outcome: FVC AUC(0-4h), Normalized by Time -- Change From Baseline to Post Dose Day 1 and Day 14
Description: as for outcome 8
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
Litres
  Day 1: number analyzed (Participants) | 39 | 34 | 37 | 40 | 40 | 40
  Day 1 | 0.158 [0.112 to 0.203] | 0.186 [0.136 to 0.235] | 0.159 [0.113 to 0.206] | 0.215 [0.171 to 0.260] | 0.036 [-0.007 to 0.079] | 0.213 [0.168 to 0.257]
  Day 14: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14 | 0.135 [0.089 to 0.181] | 0.146 [0.098 to 0.195] | 0.136 [0.089 to 0.184] | 0.194 [0.151 to 0.238] | 0.050 [0.004 to 0.095] | 0.177 [0.132 to 0.221]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.122, 95% CI 2-sided [0.058 to 0.187]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.150, 95% CI 2-sided [0.085 to 0.215]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.124, 95% CI 2-sided [0.059 to 0.189]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.180, 95% CI 2-sided [0.118 to 0.242]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.177, 95% CI 2-sided [0.115 to 0.238]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.410, ANCOVA; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.039 to 0.094]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p = 0.961, ANCOVA; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.063 to 0.066]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.070, ANCOVA; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [-0.005 to 0.119]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.454, ANCOVA; Mean Difference (Final Values) = -0.026, 95% CI 2-sided [-0.095 to 0.043]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.370, ANCOVA; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.035 to 0.095]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 11]; Test type: Superiority; p = 0.086, ANCOVA; Mean Difference (Final Values) = 0.056, 95% CI 2-sided [-0.008 to 0.120]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 12]; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Final Values) = 0.086, 95% CI 2-sided [0.020 to 0.151]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = 0.097, 95% CI 2-sided [0.029 to 0.164]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 14]; Test type: Superiority; p = 0.010, ANCOVA; Mean Difference (Final Values) = 0.087, 95% CI 2-sided [0.021 to 0.153]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.145, 95% CI 2-sided [0.081 to 0.208]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 16]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.127, 95% CI 2-sided [0.065 to 0.189]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.740, ANCOVA; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.055 to 0.078]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 18]; Test type: Superiority; p = 0.973, ANCOVA; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.064 to 0.066]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 19]; Test type: Superiority; p = 0.064, ANCOVA; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [-0.003 to 0.122]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 20]; Test type: Superiority; p = 0.774, ANCOVA; Mean Difference (Final Values) = -0.010, 95% CI 2-sided [-0.079 to 0.059]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.151, ANCOVA; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.018 to 0.113]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.076, ANCOVA; Mean Difference (Final Values) = 0.058, 95% CI 2-sided [-0.006 to 0.122]

10. Secondary Outcome: FVC Peak(0-4h), Normalized by Time -- Change From Baseline to Post Dose Day 1 and Day 14
Description: as for outcome 8
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
Litres
  Day 1 | 0.331 [0.277 to 0.384] | 0.347 [0.290 to 0.404] | 0.354 [0.299 to 0.408] | 0.367 [0.315 to 0.419] | 0.216 [0.166 to 0.267] | 0.385 [0.333 to 0.437]
  Day 14: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14 | 0.310 [0.259 to 0.361] | 0.331 [0.277 to 0.385] | 0.304 [0.251 to 0.358] | 0.350 [0.301 to 0.399] | 0.198 [0.147 to 0.250] | 0.340 [0.290 to 0.390]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = 0.114, 95% CI 2-sided [0.039 to 0.190]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.130, 95% CI 2-sided [0.055 to 0.206]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.137, 95% CI 2-sided [0.061 to 0.213]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.151, 95% CI 2-sided [0.078 to 0.223]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.168, 95% CI 2-sided [0.097 to 0.240]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.679, ANCOVA; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.061 to 0.093]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p = 0.549, ANCOVA; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.052 to 0.098]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.323, ANCOVA; Mean Difference (Final Values) = 0.036, 95% CI 2-sided [-0.036 to 0.109]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.866, ANCOVA; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.073 to 0.087]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.596, ANCOVA; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.055 to 0.096]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Test type: Superiority — Day 1 Comparison groups were: Treatment D (CHF 1531 pMDI 48 μg TDD) versus Treatment C (CHF 1531 pMDI 24 μg TDD). Statistical analysis was performed as described for the statistical analysis #1 of this outcome measure; p = 0.720, ANCOVA; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.061 to 0.088]
Statistical Analysis 12: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 12]; Test type: Superiority; p = 0.003, ANCOVA; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [0.038 to 0.185]
Statistical Analysis 13: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.133, 95% CI 2-sided [0.057 to 0.209]
Statistical Analysis 14: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 14]; Test type: Superiority; p = 0.005, ANCOVA; Mean Difference (Final Values) = 0.106, 95% CI 2-sided [0.032 to 0.180]
Statistical Analysis 15: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.152, 95% CI 2-sided [0.081 to 0.223]
Statistical Analysis 16: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 16]; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [0.072 to 0.212]
Statistical Analysis 17: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.573, ANCOVA; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [-0.053 to 0.096]
Statistical Analysis 18: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 18]; Test type: Superiority; p = 0.881, ANCOVA; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.078 to 0.067]
Statistical Analysis 19: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 19]; Test type: Superiority; p = 0.261, ANCOVA; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.030 to 0.110]
Statistical Analysis 20: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 20]; Test type: Superiority; p = 0.493, ANCOVA; Mean Difference (Final Values) = -0.027, 95% CI 2-sided [-0.104 to 0.051]
Statistical Analysis 21: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.616, ANCOVA; Mean Difference (Final Values) = 0.019, 95% CI 2-sided [-0.055 to 0.092]
Statistical Analysis 22: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.212, ANCOVA; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [-0.026 to 0.118]

11. Secondary Outcome: Pre-dose Morning FEV1 (L) -- Change From Baseline to Post Dose Day 14
Description: as for outcome 7
Time Frame: Baseline, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 35 | 40 | 37 | 41
Litres | 0.071 [0.021 to 0.120] | 0.102 [0.049 to 0.155] | 0.073 [0.021 to 0.125] | 0.149 [0.101 to 0.197] | 0.037 [-0.013 to 0.087] | 0.126 [0.077 to 0.175]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.361, ANCOVA; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.039 to 0.106]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.085, ANCOVA; Mean Difference (Final Values) = 0.065, 95% CI 2-sided [-0.009 to 0.138]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.328, ANCOVA; Mean Difference (Final Values) = 0.036, 95% CI 2-sided [-0.037 to 0.109]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [0.042 to 0.182]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.011, ANCOVA; Mean Difference (Final Values) = 0.089, 95% CI 2-sided [0.020 to 0.158]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.404, ANCOVA; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.042 to 0.104]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p = 0.942, ANCOVA; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.069 to 0.074]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.027, ANCOVA; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [0.009 to 0.147]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.463, ANCOVA; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.104 to 0.048]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.200, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [-0.025 to 0.119]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 11]; Test type: Superiority; p = 0.037, ANCOVA; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [0.005 to 0.146]

12. Secondary Outcome: Pre-dose Morning FVC -- Change From Baseline to Post Dose Day 14
Description: as for outcome 8
Time Frame: Baseline, Day 14 post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litres
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 35 | 40 | 37 | 41
Litres | 0.048 [-0.005 to 0.102] | 0.044 [-0.013 to 0.101] | 0.048 [-0.009 to 0.104] | 0.114 [0.062 to 0.166] | 0.053 [-0.000 to 0.107] | 0.114 [0.061 to 0.166]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Day 14 Comparison groups were: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). This secondary efficacy variable was analyzed using the ANCOVA model that was also used for the primary efficacy analysis, without adjusting for multiplicity; Test type: Superiority; p = 0.896, ANCOVA; Mean Difference (Final Values) = -0.005, 95% CI 2-sided [-0.083 to 0.073]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 13]; Test type: Superiority; p = 0.810, ANCOVA; Mean Difference (Final Values) = -0.010, 95% CI 2-sided [-0.089 to 0.070]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 14]; Test type: Superiority; p = 0.882, ANCOVA; Mean Difference (Final Values) = -0.006, 95% CI 2-sided [-0.084 to 0.073]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.115, ANCOVA; Mean Difference (Final Values) = 0.060, 95% CI 2-sided [-0.015 to 0.136]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 16]; Test type: Superiority; p = 0.111, ANCOVA; Mean Difference (Final Values) = 0.060, 95% CI 2-sided [-0.014 to 0.134]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 17]; Test type: Superiority; p = 0.911, ANCOVA; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.083 to 0.074]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 18]; Test type: Superiority; p = 0.985, ANCOVA; Mean Difference (Final Values) = -0.001, 95% CI 2-sided [-0.078 to 0.077]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 19]; Test type: Superiority; p = 0.084, ANCOVA; Mean Difference (Final Values) = 0.066, 95% CI 2-sided [-0.009 to 0.140]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 20]; Test type: Superiority; p = 0.928, ANCOVA; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.078 to 0.086]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 21]; Test type: Superiority; p = 0.078, ANCOVA; Mean Difference (Final Values) = 0.070, 95% CI 2-sided [-0.008 to 0.148]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.089, ANCOVA; Mean Difference (Final Values) = 0.066, 95% CI 2-sided [-0.010 to 0.143]

13. Secondary Outcome: Time to Onset of Action -- Change From Baseline in Post-dose FEV1 ≥12% and ≥200 mL to Post Dose Day 1
Description: Spirometry, used to measure FEV1, was performed according to internationally accepted standards.
  For patients receiving the same treatment twice, the analysis includes only data from the first instance of each treatment.
  Definitions:
  Time to onset of action=The time (in minutes) from receiving the study drug on Day 1, until the FEV1 change from baseline is ≥200 mL; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose) on Day 1 of the treatment period;
Time Frame: Baseline, Day 1 post-dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
minutes | 358.8 [43.1 to NA] — NA: Censoring for patients not achieving onset of action | 60.3 [31.3 to NA] — NA: Censoring for patients not achieving onset of action | 33.6 [16.0 to 118.8] | 44.3 [16.0 to 240.1] | NA [NA to NA] — NA: Censoring for patients not achieving onset of action | 45.5 [32.6 to 66.8]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Day 1 Comparison groups were: Treatment A (CHF 1531 pMDI 6 μg TDD) versus Treatment E (Placebo). Time to onset of action was analyzed using a Cox proportional hazard model stratified by patient, including treatment and period as a factor, and baseline FEV1 as covariate. For patients receiving the same treatment twice, the analysis includes only data from the first instance of each treatment; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 18.01, 95% CI 2-sided [4.25 to 76.37]
Statistical Analysis 2: Comparison: Treatment B vs Treatment E; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 31.67, 95% CI 2-sided [7.52 to 133.47]
Statistical Analysis 3: Comparison: Treatment C vs Treatment E; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 44.24, 95% CI 2-sided [10.23 to 191.34]
Statistical Analysis 4: Comparison: Treatment D vs Treatment E; [analysis description as in outcome 6, analysis 4]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 40.32, 95% CI 2-sided [9.54 to 170.45]
Statistical Analysis 5: Comparison: Treatment E vs Treatment F; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 22.91, 95% CI 2-sided [5.70 to 92.06]
Statistical Analysis 6: Comparison: Treatment A vs Treatment B; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.195, Regression, Cox; Hazard Ratio (HR) = 1.76, 95% CI 2-sided [0.75 to 4.13]
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p = 0.037, Regression, Cox; Risk Ratio (RR) = 2.46, 95% CI 2-sided [1.06 to 5.72]
Statistical Analysis 8: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.042, Regression, Cox; Hazard Ratio (HR) = 2.24, 95% CI 2-sided [1.03 to 4.86]
Statistical Analysis 9: Comparison: Treatment B vs Treatment C; [analysis description as in outcome 6, analysis 9]; Test type: Superiority; p = 0.435, Regression, Cox; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.60 to 3.23]
Statistical Analysis 10: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 6, analysis 10]; Test type: Superiority; p = 0.564, Regression, Cox; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.56 to 2.89]
Statistical Analysis 11: Comparison: Treatment C vs Treatment D; Test type: Superiority — [test comment as in outcome 10, analysis 11]; p = 0.818, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.41 to 2.01]

14. Secondary Outcome: Patients Achieving Onset of Action -- Change From Baseline in Post-dose FEV1 ≥12% and ≥200 mL to Post Dose Day 1
Description: Patients achieving onset of action, defined as a change from baseline in post-dose FEV1 ≥12% and ≥200 mL, on Day 1. These are the subjects who contributed to the results, reported as median and 95% CI for 'Time to onset of action' presented in the Outcome Measure 13, above.
  For patients receiving the same treatment twice, the analysis includes only data from the first instance of each treatment.
  Definitions:
  Onset of action=Change from baseline in post-dose FEV1 ≥12% and ≥200 mL; Baseline=Baseline value was the average of the pre-dose measurements (at 45 mins and 15 mins pre-dose);
Time Frame: Baseline, Day 1 post-dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
Participants | 23 | 22 | 30 | 29 | 11 | 31

15. Secondary Outcome: Vital Signs (Systolic Blood Pressure [SBP] and Diastolic Blood Pressure [DBP]) -- Change From Baseline for Post-dose on Day 1 and on Day 14
Description: Vital signs -- Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) were measured at pre-specified times (at baseline - pre dose and on Day 14 of each treatment period or on the day of early study termination).
  Results are shown by treatment group, as change from baseline (in mmHg).
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  Definitions:
  For safety variables, the baseline for each treatment period was defined as pre-dose measurements on Day 1 of each treatment period; Day 14=The day of the last dosing of a treatment period. Day 14 of the second, third, and fourth treatment periods (day of last dosing); treatments were separated by a 2-week wash-out interval;
Time Frame: Baseline, Day 1 and Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
mmHg
  SBP, Day 1, 30 min post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  SBP, Day 1, 30 min post-dose | -1.2 [-14 to 9] | 0.2 [-23 to 11] | -0.8 [-35 to 19] | -1.2 [-21 to 17] | -0.5 [-12 to 9] | -0.8 [-15 to 11]
  SBP, Day 1, 1 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 40
  SBP, Day 1, 1 h post-dose | -0.1 [-15 to 17] | 0.5 [-18 to 14] | -0.6 [-31 to 11] | -0.6 [-18 to 15] | -0.8 [-17 to 16] | -0.8 [-13 to 11]
  SBP, Day 1, 4 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  SBP, Day 1, 4 h post-dose | 1.7 [-11 to 20] | 0.4 [-13 to 15] | -0.9 [-32 to 16] | 0.9 [-12 to 17] | 0.2 [-14 to 17] | 0.5 [-25 to 11]
  SBP, Day 1, 8 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  SBP, Day 1, 8 h post-dose | 0.8 [-16 to 18] | 0.2 [-19 to 19] | 1.1 [-23 to 31] | 0.7 [-15 to 13] | 0.5 [-18 to 14] | 2.5 [-13 to 26]
  SBP, Day 1, 12 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  SBP, Day 1, 12 h post-dose | 1.8 [-13 to 21] | 2.1 [-17 to 18] | 3.0 [-24 to 28] | 1.4 [-11 to 18] | -0.1 [-16 to 16] | 3.4 [-12 to 28]
  SBP, Day 14, pre-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  SBP, Day 14, pre-dose | 1.0 [-15 to 15] | -1.8 [-19 to 20] | 0.0 [-17 to 23] | -0.4 [-22 to 23] | -2.5 [-19 to 22] | -0.3 [-14 to 18]
  SBP, Day 14, 30 min post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  SBP, Day 14, 30 min post-dose | 0.3 [-23 to 23] | -3.1 [-24 to 15] | -0.7 [-25 to 24] | -0.7 [-27 to 36] | -3.6 [-16 to 15] | -2.5 [-19 to 12]
  SBP, Day 14, 1 h post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  SBP, Day 14, 1 h post-dose | 0.1 [-17 to 16] | -1.8 [-29 to 25] | -1.8 [-29 to 36] | -1.9 [-29 to 33] | -1.7 [-18 to 12] | -1.1 [-14 to 17]
  SBP, Day 14, 4 h post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  SBP, Day 14, 4 h post-dose | 0.9 [-26 to 19] | 0.1 [-26 to 26] | -1.4 [-20 to 15] | 1.0 [-13 to 25] | -0.5 [-26 to 49] | -0.8 [-20 to 22]
  SBP, Day 14, 8 h post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  SBP, Day 14, 8 h post-dose | 0.7 [-20 to 23] | 1.3 [-13 to 16] | 1.1 [-20 to 25] | 0.6 [-16 to 28] | -3.3 [-27 to 27] | 0.6 [-13 to 13]
  SBP, Day 14, 12 h post-dose: number analyzed (Participants) | 35 | 34 | 31 | 36 | 30 | 41
  SBP, Day 14, 12 h post-dose | 1.2 [-18 to 17] | 1.0 [-23 to 29] | 1.5 [-26 to 26] | 4.4 [-18 to 39] | -0.3 [-20 to 43] | 2.5 [-11 to 19]
  DBP, Day 1, 30 min post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  DBP, Day 1, 30 min post-dose | -2.1 [-19 to 10] | -1.5 [-19 to 10] | -1.2 [-21 to 8] | -2.0 [-20 to 13] | -0.3 [-11 to 14] | -1.2 [-17 to 12]
  DBP, Day 1, 1 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 40
  DBP, Day 1, 1 h post-dose | 0.0 [-8 to 9] | -1.9 [-18 to 12] | -0.4 [-14 to 17] | -1.6 [-17 to 11] | -2.5 [-12 to 8] | -1.7 [-15 to 15]
  DBP, Day 1, 4 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  DBP, Day 1, 4 h post-dose | -0.6 [-11 to 9] | -1.4 [-13 to 9] | -0.4 [-11 to 14] | -1.0 [-20 to 15] | -1.6 [-13 to 8] | -1.0 [-16 to 14]
  DBP, Day 1, 8 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  DBP, Day 1, 8 h post-dose | -1.5 [-15 to 10] | -0.9 [-10 to 15] | -0.4 [-13 to 10] | -1.9 [-16 to 11] | -1.7 [-13 to 9] | 0.4 [-17 to 12]
  DBP, Day 1, 12 h post-dose: number analyzed (Participants) | 35 | 34 | 34 | 36 | 35 | 41
  DBP, Day 1, 12 h post-dose | -0.5 [-11 to 16] | -0.1 [-14 to 15] | 0.4 [-14 to 11] | -1.0 [-11 to 14] | -0.3 [-14 to 9] | 0.0 [-13 to 13]
  DBP, Day 14, pre-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  DBP, Day 14, pre-dose | -1.2 [-13 to 8] | 0.1 [-10 to 19] | 1.1 [-13 to 10] | -0.1 [-16 to 14] | -0.6 [-13 to 10] | -0.7 [-13 to 17]
  DBP, Day 14, 30 min post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  DBP, Day 14, 30 min post-dose | -0.2 [-14 to 17] | -2.1 [-21 to 20] | -0.8 [-20 to 8] | -2.9 [-20 to 16] | -1.5 [-12 to 10] | -2.0 [-14 to 14]
  DBP, Day 14, 1 h post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  DBP, Day 14, 1 h post-dose | -0.3 [-13 to 13] | -2.4 [-24 to 24] | -0.5 [-14 to 12] | -2.4 [-24 to 25] | -1.8 [-12 to 16] | -1.6 [-18 to 14]
  DBP, Day 14, 4 h post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  DBP, Day 14, 4 h post-dose | -1.0 [-15 to 9] | -1.5 [-18 to 19] | -1.7 [-12 to 9] | -2.5 [-17 to 10] | 0.4 [-12 to 24] | -2.3 [-16 to 24]
  DBP, Day 14, 8 h post-dose: number analyzed (Participants) | 35 | 34 | 32 | 36 | 31 | 41
  DBP, Day 14, 8 h post-dose | -1.1 [-15 to 15] | -1.0 [-18 to 18] | 0.3 [-11 to 13] | -2.6 [-20 to 14] | -1.7 [-19 to 15] | -1.3 [-14 to 13]
  DBP, Day 14, 12 h post-dose: number analyzed (Participants) | 35 | 34 | 31 | 36 | 30 | 41
  DBP, Day 14, 12 h post-dose | 0.0 [-11 to 18] | -0.7 [-15 to 21] | 0.7 [-10 to 13] | -0.6 [-19 to 14] | 1.4 [-15 to 25] | -0.1 [-10 to 14]

16. Secondary Outcome: 12-lead ECG Parameter -- Heart Rate (HR) -- Change From Baseline Post-dose to Post Dose Day 1 and Day 14
Description: Results are shown by treatment group, as change from baseline (in bpm).
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  For safety variables, the baseline for each period was defined as pre-dose measurements on Day 1 of each treatment period.
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (Full Range); unit: bpm
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
bpm
  Day 1, 30 min post-dose | 0.3 [-14 to 23] | 1.2 [-11 to 21] | 1.7 [-7 to 22] | 2.5 [-10 to 15] | -2.4 [-21 to 15] | -0.3 [-20 to 13]
  Day 1, 1h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 40
  Day 1, 1h post-dose | -1.3 [-15 to 15] | 0.3 [-17 to 20] | 2.7 [-9 to 18] | 1.5 [-11 to 13] | -1.8 [-22 to 13] | -1.2 [-18 to 15]
  Day 1, 4h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 39 | 40 | 40
  Day 1, 4h post-dose | 2.1 [-12 to 14] | 1.5 [-19 to 16] | 3.3 [-10 to 15] | 5.3 [-10 to 21] | 0.2 [-17 to 19] | 3.2 [-16 to 27]
  Day 1, 8h post-dose | 5.0 [-19 to 27] | 2.4 [-16 to 21] | 5.0 [-8 to 15] | 3.9 [-12 to 23] | 0.5 [-21 to 18] | 2.1 [-18 to 23]
  Day 1, 12h post-dose | 5.1 [-13 to 28] | 5.5 [-13 to 32] | 5.5 [-15 to 24] | 7.6 [-12 to 28] | 2.4 [-18 to 25] | 5.2 [-15 to 24]
  Day 14, pre-dose: number analyzed (Participants) | 39 | 35 | 35 | 40 | 37 | 41
  Day 14, pre-dose | 2.5 [-14 to 22] | 0.1 [-13 to 13] | 3.1 [-6 to 17] | 2.0 [-12 to 16] | 0.7 [-26 to 15] | 0.4 [-11 to 16]
  Day 14, 30 min post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 30 min post-dose | 2.9 [-12 to 25] | -0.8 [-21 to 18] | 1.6 [-9 to 12] | 4.3 [-10 to 20] | -1.5 [-28 to 19] | 1.3 [-19 to 32]
  Day 14, 1h post-dose: number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  Day 14, 1h post-dose | 1.9 [-16 to 26] | -1.2 [-18 to 15] | 1.6 [-11 to 12] | 3.2 [-12 to 19] | -1.2 [-31 to 29] | 0.4 [-22 to 30]
  Day 14, 4h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 4h post-dose | 2.8 [-14 to 24] | 2.3 [-19 to 14] | 6.7 [-7 to 25] | 3.4 [-14 to 19] | 1.8 [-22 to 15] | 2.3 [-25 to 19]
  Day 14, 8h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 8h post-dose | 5.5 [-16 to 26] | 3.5 [-22 to 19] | 4.9 [-16 to 19] | 3.8 [-12 to 24] | 1.6 [-21 to 23] | 2.6 [-22 to 22]
  Day 14, 12h post-dose: number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
  Day 14, 12h post-dose | 7.4 [-17 to 34] | 7.5 [-17 to 30] | 6.7 [-15 to 19] | 5.4 [-16 to 27] | 0.5 [-23 to 16] | 5.1 [-19 to 30]

17. Secondary Outcome: Heart Rate (HR) AUC(0-4h), Normalized by Time -- Change From Baseline Post-dose to Post Dose Day 1 and Day 14
Description: Heart rate HR AUC(0-4h) normalized by time. Results are shown by treatment group, as change from baseline (in bpm).
  The HR AUC(0-4h) normalized by time is calculated based on the actual times, using the linear trapezoidal rule.
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  For safety variables, the baseline for each period was defined as pre-dose measurements on Day 1 of each treatment period.
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (90% Confidence Interval); unit: bpm
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
bpm
  Day 1: number analyzed (Participants) | 39 | 35 | 37 | 39 | 40 | 39
  Day 1 | 0.2 [-0.9 to 1.3] | 0.8 [-1.0 to 2.6] | 2.7 [1.4 to 4.0] | 3.0 [1.7 to 4.2] | -1.0 [-2.8 to 0.7] | 0.3 [-1.2 to 1.7]
  Day 14: number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  Day 14 | 2.3 [0.3 to 4.3] | 0.2 [-1.7 to 2.2] | 3.5 [1.9 to 5.1] | 3.3 [1.4 to 5.3] | -0.1 [-2.5 to 2.2] | 1.2 [-0.9 to 3.3]

18. Secondary Outcome: Heart Rate (HR) Peak(0-4h), Normalized by Time -- Change From Baseline Post-dose to Post Dose Day 1 and Day 14
Description: Heart rate (HR) peak(0-4h) normalized by time.
  Results are shown by treatment group, as change from baseline (in bpm).
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  For safety variables, the baseline for each period was defined as pre-dose measurements on Day 1 of each treatment period.
  Definitions:
  HR=Heart rate; HR peak(0-4h)=The maximum observed value over 4 hours following dosing;
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (90% Confidence Interval); unit: bpm
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
bpm
  Day 1: number analyzed (Participants) | 39 | 35 | 37 | 39 | 40 | 39
  Day 1 | 4.7 [3.1 to 6.2] | 4.4 [2.2 to 6.6] | 6.5 [4.7 to 8.3] | 7.5 [5.9 to 9.0] | 2.9 [0.8 to 5.0] | 5.1 [3.3 to 6.9]
  Day 14: number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  Day 14 | 6.1 [3.8 to 8.5] | 4.8 [2.5 to 7.1] | 8.3 [6.2 to 10.3] | 7.3 [5.4 to 9.2] | 4.4 [1.6 to 7.1] | 5.2 [2.9 to 7.5]

19. Secondary Outcome: Heart Rate (HR) AUC(0-4h) and Peak(0-4h), Normalized by Time -- Change From Pre-dose to Post Dose Day 14
Description: Heart rate (HR) AUC(0-4h) and HR peak(0-4h), normalized by time (in bpm).
  Results are shown as change from pre-dose on Day 14 (in bpm).
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  Definitions:
  HR=Heart rate; HR AUC(0-4h)=Area under the curve between 0 and 4 h for heart rate; HR peak(0-4h)=The maximum observed value over 4 h after dosing;
Time Frame: Baseline, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (90% Confidence Interval); unit: bpm
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
bpm
  HR AUC(0-4h): number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  HR AUC(0-4h) | -0.4 [-1.7 to 1.0] | 0.5 [-1.0 to 2.1] | 0.4 [-0.9 to 1.7] | 1.3 [-0.1 to 2.7] | -0.2 [-1.7 to 1.3] | 0.9 [-0.6 to 2.3]
  HR peak(0-4h): number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  HR peak(0-4h) | 3.5 [1.6 to 5.4] | 5.1 [3.2 to 6.9] | 5.1 [3.3 to 6.9] | 5.3 [3.8 to 6.7] | 4.3 [2.3 to 6.2] | 4.8 [3.1 to 6.6]

20. Secondary Outcome: 12-lead Electrocardiogram (ECG) Parameter (QTcF Interval) -- Change From Baseline Post-dose to Post Dose Day 1 and Day 14
Description: 12-lead electrocardiogram (ECG) parameters were monitored during the study. Results are shown by treatment group, as change from baseline (in msec).
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  For safety variables, the baseline for each period was defined as pre-dose measurements on Day 1 of each treatment period.
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (Full Range); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
msec
  Day 1, 30 min post-dose | 3.9 [-28 to 29] | 3.8 [-5 to 29] | 2.7 [-22 to 23] | 4.9 [-27 to 24] | -0.2 [-30 to 25] | 1.4 [-27 to 67]
  Day 1, 1h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 40
  Day 1, 1h post-dose | 2.1 [-44 to 19] | 1.4 [-29 to 27] | 3.9 [-16 to 25] | 4.2 [-21 to 31] | 0.4 [-55 to 26] | -0.9 [-24 to 28]
  Day 1, 4h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 39 | 40 | 40
  Day 1, 4h post-dose | 2.5 [-39 to 24] | 1.5 [-30 to 25] | 0.8 [-28 to 28] | 2.4 [-17 to 22] | -2.4 [-42 to 16] | -1.3 [-30 to 16]
  Day 1, 8h post-dose | 2.4 [-25 to 15] | 1.1 [-14 to 31] | 0.6 [-27 to 24] | 0.8 [-18 to 23] | -0.2 [-20 to 25] | -2.4 [-37 to 19]
  Day 1, 12h post-dose | 2.0 [-26 to 25] | 0.9 [-21 to 32] | -0.3 [-25 to 21] | 1.1 [-21 to 33] | -1.5 [-25 to 30] | -2.2 [-44 to 20]
  Day 14, pre-dose: number analyzed (Participants) | 39 | 35 | 35 | 40 | 37 | 41
  Day 14, pre-dose | 1.5 [-26 to 30] | -0.4 [-30 to 33] | 1.6 [-20 to 28] | 5.8 [-22 to 68] | -2.3 [-17 to 27] | 1.2 [-46 to 29]
  Day 14, 30 min post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 30 min post-dose | 4.4 [-28 to 30] | 1.0 [-29 to 37] | 3.5 [-28 to 31] | 10.4 [-23 to 41] | 1.9 [-29 to 22] | 1.7 [-29 to 29]
  Day 14, 1h post-dose: number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  Day 14, 1h post-dose | 4.0 [-19 to 23] | 1.0 [-45 to 37] | 1.9 [-32 to 31] | 7.7 [-25 to 44] | 0.9 [-44 to 28] | 0.6 [-36 to 29]
  Day 14, 4h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 4h post-dose | 3.8 [-9 to 29] | 0.9 [-26 to 37] | 1.1 [-33 to 30] | 5.0 [-37 to 40] | -1.1 [-28 to 28] | -1.1 [-48 to 25]
  Day 14, 8h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 8h post-dose | 3.4 [-21 to 30] | 1.7 [-23 to 29] | 1.7 [-35 to 28] | 2.2 [-37 to 44] | 1.5 [-28 to 34] | 0.4 [-38 to 30]
  Day 14, 12h post-dose: number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
  Day 14, 12h post-dose | 3.7 [-15 to 29] | 1.7 [-21 to 25] | -0.9 [-20 to 32] | 3.7 [-17 to 34] | -0.6 [-22 to 20] | -1.6 [-36 to 29]

21. Secondary Outcome: 12-lead Electrocardiogram (ECG) Parameter (PR Interval) -- Change From Baseline Post-dose to Post Dose Day 1 and Day 14
Description: as for outcome 20
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (Full Range); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
msec
  Day 1, 30 min post-dose | -0.1 [-33 to 22] | 1.6 [-12 to 18] | -1.3 [-10 to 9] | -3.6 [-71 to 15] | 1.0 [-13 to 15] | 3.2 [-11 to 24]
  Day 1, 1h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 40
  Day 1, 1h post-dose | 1.1 [-13 to 16] | 2.2 [-16 to 21] | -1.1 [-27 to 17] | -0.7 [-66 to 13] | 0.4 [-13 to 18] | 2.0 [-11 to 20]
  Day 1, 4h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 39 | 40 | 40
  Day 1, 4h post-dose | -1.2 [-14 to 11] | 1.6 [-17 to 24] | -1.5 [-16 to 16] | -4.0 [-88 to 14] | -1.6 [-33 to 21] | 1.9 [-13 to 37]
  Day 1, 8h post-dose | -1.9 [-16 to 23] | -0.5 [-14 to 20] | -3.0 [-16 to 10] | -2.6 [-74 to 10] | -2.4 [-29 to 16] | -0.0 [-13 to 27]
  Day 1, 12h post-dose | -3.4 [-17 to 14] | -2.3 [-18 to 18] | -3.8 [-15 to 17] | -3.0 [-46 to 28] | -2.6 [-15 to 19] | -1.7 [-14 to 21]
  Day 14, pre-dose: number analyzed (Participants) | 39 | 35 | 35 | 40 | 37 | 41
  Day 14, pre-dose | 1.3 [-16 to 23] | 3.7 [-17 to 25] | -1.7 [-22 to 15] | -2.9 [-53 to 18] | 0.1 [-13 to 15] | 2.2 [-15 to 28]
  Day 14, 30 min post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 30 min post-dose | -0.2 [-24 to 22] | 4.5 [-12 to 27] | -1.5 [-20 to 17] | -3.1 [-85 to 19] | 3.4 [-15 to 26] | 5.1 [-19 to 67]
  Day 14, 1h post-dose: number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  Day 14, 1h post-dose | 1.0 [-24 to 30] | 5.7 [-13 to 35] | 0.1 [-19 to 25] | -1.6 [-93 to 19] | 5.2 [-8 to 67] | 6.1 [-14 to 62]
  Day 14, 4h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 4h post-dose | -1.5 [-28 to 14] | 2.5 [-11 to 23] | -2.5 [-22 to 14] | -3.2 [-76 to 21] | 0.8 [-18 to 20] | 1.3 [-33 to 29]
  Day 14, 8h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 8h post-dose | -2.6 [-32 to 17] | 1.5 [-13 to 46] | -3.2 [-25 to 22] | -5.4 [-71 to 8] | -1.1 [-20 to 16] | 0.8 [-28 to 23]
  Day 14, 12h post-dose: number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
  Day 14, 12h post-dose | -5.0 [-40 to 11] | 1.7 [-22 to 59] | -4.8 [-24 to 19] | -1.4 [-27 to 27] | 0.1 [-20 to 34] | -0.3 [-18 to 19]

22. Secondary Outcome: 12-lead Electrocardiogram (ECG) Parameter (QRS Interval) -- Change From Baseline Post-dose to Post Dose Day 1 and Day 14
Description: as for outcome 20
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (Full Range); unit: msec
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
msec
  Day 1, 30 min post-dose | 1.2 [-9 to 9] | 1.2 [-8 to 11] | 1.7 [-6 to 8] | 1.1 [-8 to 10] | 0.8 [-7 to 7] | 1.3 [-7 to 7]
  Day 1, 1h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 40
  Day 1, 1h post-dose | 1.3 [-7 to 11] | 1.0 [-9 to 11] | 1.2 [-6 to 13] | 1.6 [-8 to 13] | 1.0 [-5 to 8] | 1.4 [-6 to 8]
  Day 1, 4h post-dose: number analyzed (Participants) | 39 | 35 | 37 | 39 | 40 | 40
  Day 1, 4h post-dose | 1.2 [-6 to 13] | 2.1 [-11 to 14] | 2.2 [-6 to 18] | 2.1 [-6 to 12] | 1.0 [-6 to 11] | 1.1 [-6 to 12]
  Day 1, 8h post-dose | 0.6 [-9 to 9] | 0.9 [-8 to 10] | 1.3 [-6 to 13] | 0.5 [-9 to 11] | -0.2 [-9 to 10] | 0.5 [-10 to 8]
  Day 1, 12h post-dose | 0.5 [-9 to 12] | 1.0 [-13 to 8] | 1.0 [-9 to 10] | 0.9 [-9 to 9] | 0.4 [-9 to 8] | 0.8 [-8 to 7]
  Day 14, pre-dose: number analyzed (Participants) | 39 | 35 | 35 | 40 | 37 | 41
  Day 14, pre-dose | 0.5 [-9 to 13] | 1.0 [-12 to 10] | -0.5 [-10 to 10] | 1.7 [-8 to 17] | -0.9 [-12 to 7] | 0.8 [-8 to 8]
  Day 14, 30 min post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 30 min post-dose | 1.4 [-7 to 14] | 1.6 [-10 to 12] | 0.5 [-7 to 11] | 2.4 [-5 to 12] | -0.3 [-8 to 11] | 1.7 [-6 to 9]
  Day 14, 1h post-dose: number analyzed (Participants) | 38 | 34 | 35 | 40 | 35 | 41
  Day 14, 1h post-dose | 1.3 [-5 to 15] | 0.9 [-10 to 11] | 0.4 [-7 to 9] | 2.3 [-9 to 11] | 0.0 [-12 to 13] | 1.0 [-10 to 9]
  Day 14, 4h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 4h post-dose | 2.0 [-10 to 15] | 1.8 [-9 to 19] | 0.6 [-7 to 9] | 2.8 [-11 to 12] | -0.2 [-9 to 8] | 1.1 [-6 to 11]
  Day 14, 8h post-dose: number analyzed (Participants) | 38 | 35 | 35 | 40 | 36 | 41
  Day 14, 8h post-dose | 0.7 [-11 to 15] | 1.2 [-10 to 12] | 0.1 [-11 to 12] | 1.4 [-7 to 10] | -0.8 [-10 to 9] | 0.9 [-12 to 12]
  Day 14, 12h post-dose: number analyzed (Participants) | 38 | 35 | 34 | 40 | 35 | 41
  Day 14, 12h post-dose | 0.8 [-8 to 15] | 0.4 [-13 to 10] | 0.3 [-9 to 11] | 1.4 [-6 to 17] | -1.0 [-9 to 8] | 0.5 [-10 to 14]

23. Secondary Outcome: Serum Potassium -- Change From Baseline Post-dose to Post Dose Day 1 and Day 14
Description: Serum potassium level was monitored during the study. Results are shown by treatment group, as change from baseline (in mmol/L).
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  For safety variables, the baseline for each period was defined as pre-dose measurements on Day 1 of each treatment period.
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
mmol/L
  Day 1; 1.5h post-dose: number analyzed (Participants) | 35 | 33 | 32 | 35 | 34 | 40
  Day 1; 1.5h post-dose | -0.01 [-0.9 to 0.8] | -0.05 [-1.1 to 0.7] | -0.08 [-1.2 to 0.6] | -0.17 [-0.7 to 0.3] | -0.06 [-0.9 to 0.6] | -0.18 [-1.0 to 0.6]
  Day 1; 3h post-dose: number analyzed (Participants) | 34 | 33 | 32 | 35 | 34 | 40
  Day 1; 3h post-dose | -0.06 [-0.9 to 1.0] | -0.08 [-0.8 to 0.5] | -0.23 [-1.3 to 0.3] | -0.28 [-1.5 to 0.4] | 0.03 [-0.7 to 0.9] | -0.21 [-1.0 to 0.9]
  Day 1; 5h post-dose: number analyzed (Participants) | 35 | 34 | 32 | 35 | 34 | 40
  Day 1; 5h post-dose | -0.14 [-0.6 to 0.5] | -0.03 [-0.6 to 1.2] | -0.12 [-1.0 to 0.6] | -0.19 [-1.6 to 1.0] | -0.04 [-0.9 to 0.5] | -0.20 [-1.3 to 0.5]
  Day 1; 7h post-dose: number analyzed (Participants) | 34 | 32 | 31 | 35 | 35 | 40
  Day 1; 7h post-dose | -0.02 [-0.6 to 0.8] | -0.00 [-0.9 to 0.7] | -0.05 [-0.8 to 0.8] | -0.16 [-1.8 to 0.6] | 0.04 [-0.7 to 0.9] | -0.14 [-1.4 to 1.0]
  Day 1; 11h post-dose: number analyzed (Participants) | 35 | 32 | 32 | 33 | 32 | 39
  Day 1; 11h post-dose | 0.07 [-0.7 to 1.0] | 0.02 [-0.5 to 1.1] | -0.08 [-1.2 to 0.9] | -0.10 [-0.8 to 0.7] | 0.01 [-1.0 to 0.6] | -0.13 [-1.4 to 0.7]
  Day 14; pre-dose: number analyzed (Participants) | 35 | 34 | 31 | 35 | 30 | 40
  Day 14; pre-dose | 0.06 [-1.1 to 0.9] | -0.02 [-1.2 to 0.4] | 0.08 [-0.9 to 0.9] | -0.14 [-1.5 to 1.3] | 0.05 [-0.5 to 1.4] | -0.13 [-0.9 to 0.8]
  Day 14; 1.5h post-dose: number analyzed (Participants) | 35 | 33 | 31 | 35 | 30 | 41
  Day 14; 1.5h post-dose | -0.02 [-0.7 to 1.5] | -0.03 [-1.0 to 1.2] | -0.10 [-1.0 to 0.9] | -0.23 [-1.7 to 1.0] | -0.03 [-0.7 to 1.7] | -0.15 [-1.0 to 1.1]
  Day 14; 3h post-dose: number analyzed (Participants) | 34 | 33 | 31 | 35 | 30 | 41
  Day 14; 3h post-dose | -0.04 [-0.6 to 0.6] | -0.09 [-1.0 to 0.7] | -0.13 [-0.9 to 0.6] | -0.24 [-1.9 to 0.6] | -0.00 [-0.6 to 1.7] | -0.15 [-1.0 to 0.6]
  Day 14; 5h post-dose: number analyzed (Participants) | 34 | 34 | 30 | 35 | 29 | 40
  Day 14; 5h post-dose | -0.02 [-0.8 to 1.0] | -0.05 [-1.1 to 1.7] | -0.01 [-1.2 to 0.8] | -0.26 [-1.9 to 0.5] | 0.00 [-0.6 to 1.5] | -0.15 [-1.1 to 0.8]
  Day 14; 7h post-dose: number analyzed (Participants) | 33 | 34 | 31 | 35 | 29 | 41
  Day 14; 7h post-dose | 0.05 [-0.5 to 1.4] | 0.06 [-0.8 to 1.2] | 0.09 [-0.9 to 1.1] | -0.19 [-1.5 to 0.5] | 0.02 [-0.7 to 1.3] | -0.09 [-1.1 to 1.0]
  Day 14; 11h post-dose: number analyzed (Participants) | 34 | 32 | 31 | 35 | 28 | 40
  Day 14; 11h post-dose | 0.11 [-0.4 to 1.3] | 0.05 [-1.3 to 1.1] | 0.03 [-1.0 to 1.1] | -0.06 [-1.4 to 1.2] | 0.01 [-1.0 to 1.0] | -0.02 [-1.1 to 1.2]

24. Secondary Outcome: Serum Glucose -- Change From Baseline to Post-dose Day 1 and Day 14
Description: Serum glucose level was monitored during the study. Results are shown by treatment group, as change from baseline (in mmol/L).
  For patients receiving the same treatment in 2 periods, the average of the 2 available data points was considered in the calculation.
  For safety variables, the baseline for each period was defined as pre-dose measurements on Day 1 of each treatment period.
Time Frame: Baseline, Day 1, Day 14 post-dose
Population: Safety population:
  All randomized patients who received at least one dose of study treatment within the given period.
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 39 | 35 | 37 | 40 | 40 | 41
mmol/L
  Day 1; 1.5h post-dose: number analyzed (Participants) | 35 | 33 | 32 | 35 | 35 | 40
  Day 1; 1.5h post-dose | 0.49 [-3.0 to 5.3] | 0.34 [-4.9 to 11.7] | 0.57 [-1.7 to 6.2] | 1.19 [-1.2 to 8.4] | 0.47 [-2.0 to 4.7] | -0.06 [-7.5 to 3.6]
  Day 1; 3h post-dose: number analyzed (Participants) | 34 | 33 | 32 | 35 | 34 | 41
  Day 1; 3h post-dose | 0.45 [-3.3 to 4.8] | 0.54 [-6.0 to 13.9] | 1.10 [-2.1 to 4.8] | 1.79 [-2.2 to 5.7] | 0.26 [-3.1 to 6.6] | 0.39 [-7.2 to 4.6]
  Day 1; 5h post-dose: number analyzed (Participants) | 34 | 34 | 32 | 35 | 35 | 41
  Day 1; 5h post-dose | 0.83 [-3.2 to 6.4] | 1.12 [-3.6 to 20.5] | 1.11 [-1.0 to 4.2] | 1.58 [-1.2 to 7.6] | 0.51 [-5.1 to 10.9] | 0.44 [-1.6 to 6.3]
  Day 1; 7h post-dose: number analyzed (Participants) | 34 | 32 | 31 | 35 | 35 | 41
  Day 1; 7h post-dose | 0.81 [-2.6 to 4.8] | 0.42 [-4.7 to 5.8] | 1.24 [-1.3 to 6.5] | 1.37 [-1.6 to 8.1] | 0.84 [-1.6 to 10.4] | 0.61 [-1.2 to 8.0]
  Day 1; 11h post-dose: number analyzed (Participants) | 35 | 32 | 32 | 33 | 32 | 40
  Day 1; 11h post-dose | 0.98 [-4.1 to 6.4] | 1.08 [-3.6 to 16.1] | 1.89 [-1.6 to 6.5] | 1.42 [-2.2 to 8.7] | 1.40 [-1.1 to 6.7] | 0.90 [-2.3 to 5.2]
  Day 14; pre-dose: number analyzed (Participants) | 35 | 33 | 31 | 35 | 30 | 40
  Day 14; pre-dose | -0.34 [-8.7 to 2.9] | 0.00 [-3.8 to 2.9] | 0.49 [-0.7 to 3.3] | 0.49 [-0.8 to 10.0] | 0.37 [-0.6 to 4.1] | -0.03 [-2.8 to 2.6]
  Day 14; 1.5h post-dose: number analyzed (Participants) | 35 | 33 | 31 | 35 | 30 | 41
  Day 14; 1.5h post-dose | 0.09 [-7.0 to 9.5] | 0.26 [-3.3 to 5.1] | 0.97 [-1.3 to 4.8] | 1.21 [-0.8 to 8.9] | 0.35 [-2.0 to 3.2] | -0.03 [-4.8 to 3.9]
  Day 14; 3h post-dose: number analyzed (Participants) | 34 | 33 | 31 | 35 | 30 | 41
  Day 14; 3h post-dose | 0.09 [-10.9 to 6.3] | 0.77 [-2.1 to 4.5] | 1.31 [-1.1 to 6.0] | 1.51 [-1.7 to 9.9] | 0.25 [-2.4 to 2.7] | 0.16 [-7.0 to 4.3]
  Day 14; 5h post-dose: number analyzed (Participants) | 35 | 34 | 30 | 35 | 29 | 40
  Day 14; 5h post-dose | 0.04 [-10.8 to 5.9] | 0.90 [-1.7 to 5.4] | 1.12 [-1.9 to 4.7] | 1.16 [-1.3 to 6.7] | 0.32 [-1.8 to 4.4] | 0.53 [-3.4 to 7.2]
  Day 14; 7h post-dose: number analyzed (Participants) | 34 | 34 | 31 | 35 | 29 | 41
  Day 14; 7h post-dose | -0.04 [-9.4 to 3.4] | 0.60 [-2.5 to 7.6] | 0.73 [-1.7 to 4.3] | 1.09 [-0.7 to 12.0] | 0.25 [-6.7 to 2.4] | 0.18 [-4.6 to 2.6]
  Day 14; 11h post-dose: number analyzed (Participants) | 34 | 32 | 31 | 35 | 28 | 41
  Day 14; 11h post-dose | 0.39 [-7.9 to 5.0] | 1.30 [-1.3 to 14.1] | 1.50 [-0.5 to 5.8] | 1.47 [-1.1 to 8.9] | 1.03 [-2.7 to 3.8] | 0.68 [-2.5 to 4.8]

ADVERSE EVENTS:
Time Frame: From the first intake of study medication (Visit 2, Week 0) until study completion (Visit 10, Week 15) or study discontinuation.
Description: Safety population was used for the evaluation of treatment-emergent adverse event (TEAEs).
  The safety population is defined as all randomized patients who received at least one dose of study treatment within the given treatment period.
Groups:
- Treatment A: Treatment A CHF 1531 pMDI: 6 μg TDD
- Treatment B: Treatment B CHF 1531 pMDI: 12 μg TDD
- Treatment C: Treatment C CHF 1531 pMDI: 24 μg TDD
- Treatment D: Treatment D CHF 1531 pMDI: 48 μg TDD
- Treatment E: Treatment E Matched placebo
- Treatment F: Treatment F Formoterol fumarate IS Perforomist®: 40 μg TDD
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/36 | 0/40 | 0/44 | 0/45 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/36 | 0/40 | 0/44 | 0/45 | 0/41
Other Adverse Events (participants affected / at risk) | 2/43 | 1/36 | 2/40 | 2/44 | 0/45 | 1/41
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=43) | Treatment B (N=36) | Treatment C (N=40) | Treatment D (N=44) | Treatment E (N=45) | Treatment F (N=41)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi can publish and/or present any results of this study at scientific meetings, and to submit the clinical trial data to national and international Regulatory Authorities. Chiesi reserves the right to use such data for industrial purposes. Investigators will inform Chiesi before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT03086460/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT03086460/SAP_001.pdf